

# STATISTICAL ANALYSIS PLAN

Study CRO-PK-20-343 - Sponsor code CHL.3-01-2020

# A Phase I/II, randomized, placebo-controlled, double-masked, efficacy, safety and local tolerability study of Chloroprocaine 3% gel eye drops in healthy volunteers

Single dose, randomised, placebo-controlled, parallel-group, double-masked, efficacy, safety and local tolerability study

Test investigational product: Chloroprocaine 3% ocular gel (30 mg/mL), Sintetica S.A.,

Switzerland

Control: Placebo, vehicle for chloroprocaine 3% ocular gel,

Sintetica S.A., Switzerland

Sponsor: Sintetica S.A., Via Penate 5, 6850 Mendrisio, Switzerland

Phone: +41.91.6404250 Fax: +41.91.6468561

Investigator: Milko Radicioni, MD - Principal investigator

CROSS Research S.A., Phase I Unit

Via F.A. Giorgioli 14 CH-6864 Arzo, Switzerland Phone: +41.91.64.04.450 Fax: +41.91.64.04.451 Email: clinic@croalliance.com

Development phase: Phase I/II

Version and date: Final version 1.0, 20NOV2020

This study will be conducted in accordance with current version of Good Clinical Practice (GCP), ICH topic E6 (R2)

Property of the sponsor

May not be used, divulged, published or otherwise disclosed without the consent of the sponsor

This document comprises 30 pages plus appendices





# **VERSIONS' HISTORY**

| Version | Date of Issue | Reason for change |
|---|---|---|
| Draft version 0.1 | 12NOV2020 | Francesca Morano issued the first draft |
| Final version 1.0 | 20NOV2020 | Francesca Morano issued the final version after Blind Review Meeting |



# APPROVAL AND ACKNOWLEDGEMENT

| <b>SPONSOR</b> Sintetica S.A., Swi | tzerland | |
|---|---|---|
| | ntative (for approval and acknowledgement Clinical Development Project Manager | nt) |
| Date | Signature | |





| CRO<br>CROSS Research | S.A., Switzerland |
|---|---|
| • | epresentative (for approval and acknowledgement)<br>, Junior Biostatistician and Data Manager |
| Date | Signature |
| | Team Representative (for approval and acknowledgement) inical Projects Unit Head |
| Date | Signature |
| , | acknowledgement only) Clinical Project Leader and Senior CRA |
| Date | Signature |



# STUDY SCHEDULE

| ACTIVITIES | Screening | Intervention and assessments | Telephone call | Follow-up/ETV <sup>5</sup> |
|---|---|---|---|---|
| Visit | V1 | V2 | V3 | V4 |
| . 5555 | Day -21 / -1 | Day 1 | Day 2 | Day 7±1 |
| Informed consent | Х | · | • | Ţ. |
| Demography | X | | | |
| Ocular medical and surgical history | X | | | |
| Other medical and surgical history | X | | | |
| Physical examination | X | | | X |
| Previous medications | X | | | |
| Concomitant medications | X | X | X | X |
| Height | Х | | | |
| Body Weight | Х | | | |
| Body mass index | X | | | |
| Alcohol test | | X | | |
| Vital signs (blood pressure, heart rate) check <sup>1</sup> | X | X | | X |
| Urine pregnancy test (women) | X | | | |
| Ocular symptoms (0-100 mm VAS) <sup>1,2</sup> | Х | Х | | Х |
| Slit lamp examination <sup>1,2</sup> | Х | X | | X |
| Corneal fluorescein staining <sup>2</sup> | Х | | | X |
| Intraocular pressure <sup>2</sup> | Х | | | X |
| Fundus ophthalmology <sup>2</sup> | Х | | | X |
| Visual acuity (EDTRS) <sup>2</sup> | X | | | X |
| Inclusion / exclusion criteria check | X | X | | |
| Subject eligibility | X | X | | |
| Enrolment and randomisation | | X | | |
| Investigational product administration <sup>3</sup> | | X | | |
| Conjunctival pinching <sup>4</sup> | | X | | |
| Adverse events monitoring <sup>6</sup> | X | X | X | X |

- 1. At screening, on day 1 at pre-dose and at the end of the study day, and at follow-up/ETV
- 2. Both eyes
- 3. On day 1, after pre-dose (baseline) assessments
- 4. Study eye (right eye) only On day 1, at 20, 40 and 60 seconds and then at 5-min intervals up to 60 min post-dose, as applicable (please refer to CSP main text).
- 5. Early termination visit (ETV) in case of premature discontinuation
- 6. AEs monitored starting at the screening visit, immediately after informed consent, up to the follow-up visit/ETV.



# TABLES OF CONTENTS

| | STATISTICAL ANALYSIS PLAN | 1 |
|---|---|---|
| | VERSIONS' HISTORY | 2 |
| | APPROVAL AND ACKNOWLEDGEMENT | 3 |
| | STUDY SCHEDULE | 5 |
| | TABLES OF CONTENTS | 6 |
| | ABBREVIATIONS | 8 |
| 1 | INTRODUCTION | 9 |
| 1.1 | Changes with respect to the study protocol and its amendment(s) | 9 |
| 2 | STUDY/INVESTIGATON OBJECTIVES | 10 |
| 2.1 | Primary end-point | 10 |
| 2.2 | Secondary end-points | 10 |
| 3 | INVESTIGATIONAL PLAN | 11 |
| 3.1 | Overall study design | 11 |
| 3.2 | Discussion of design | 11 |
| 4 | STUDY POPULATION | 12 |
| 4.1 | Target population | 12 |
| 4.2 | Inclusion criteria | 12 |
| 4.3 | Exclusion criteria | 12 |
| 4.3.1 | Not allowed treatments | 13 |
| 5 | STUDY SCHEDULE | 14 |
| 5.1 | Study visits and procedures | 14 |
| 5.2 | Diet and lifestyle | 16 |
| 6 | STUDY SUBJECT IDENTIFICATION METHOD AND TREATMENT ASSIGNMENT METHOD | 17 |
| 6.1 | Unique subject identifier | 17 |
| 6.2 | Subject identifier for the study | 17 |
| 6.3 | Randomisation | 17 |
| 6.4 | Treatment allocation | 17 |
| 6.5 | Blinding | 17 |
| 6.5.1 | Emergency code and unblinding procedures | 18 |
| 6.5.2 | Emergency individual envelopes | 18 |
| 7 | STUDY EVALUATION PARAMETERS | 19 |
| 7.1 | Study variables | 19 |
| 7.1.1 | Primary variables | 19 |
| 7.1.2 | Secondary variables | 19 |
| 7.2 | Safety assessments | 19 |
| 8 | DATA MONITORING COMMITTEE AND BLIND REVIEW MEETING | 20 |
| 8.1 | Composition of data monitoring committee | 20 |
| 8.2 | Purpose and scope of the blind review meeting | 20 |
| 9 | STATISTICAL METHOD | 21 |
| 9.1 | Tables, listings and figures layout | 21 |
| 9.2 | <b>Analysis sets</b> | 21 |
| 9.2.1 | Definitions | 21 |
| 9.2.2 | Reasons for exclusion from the Full Analysis Set | 22 |
| 9.2.3 | Reasons for exclusion from the Per Protocol Set | 23 |





| 9.2.4 | Reasons for exclusion from the Safety Set | 23 |
|--------|--------------------------------------------------------|----|
| 9.3 | Sample size and power considerations | 23 |
| 9.4 | Demographic, baseline and background characteristics | 24 |
| 9.4.1 | Subjects' disposition | 24 |
| 9.4.2 | Analysis sets | 24 |
| 9.4.3 | Subjects excluded from efficacy and/or safety analysis | 24 |
| 9.4.4 | Discontinued subjects | 24 |
| 9.4.5 | Protocol deviations | 24 |
| 9.4.6 | Treatment mismatch | 24 |
| 9.4.7 | Demography | 24 |
| 9.4.8 | Inclusion/exclusion criteria not met | 25 |
| 9.4.9 | Medical and surgical history | 25 |
| 9.4.10 | Prior and concomitant medication | 25 |
| 9.4.11 | Subjects' study visits | 25 |
| 9.4.12 | Fertility status and contraceptive method | 25 |
| 9.4.13 | Alcohol breath test and pregnancy test | 25 |
| 9.5 | IMP administration | 25 |
| 9.6 | Interim analyses | 25 |
| 9.7 | Efficacy analysis | 25 |
| 9.7.1 | Primary efficacy analysis | 25 |
| 9.7.2 | Sensitivity analyses | 26 |
| 9.7.3 | Secondary efficacy analysis | 26 |
| 9.8 | Safety and tolerability analysis | 26 |
| 9.8.1 | Adverse events | 26 |
| 9.8.2 | Vital signs | 27 |
| 9.8.3 | Physical examination | 27 |
| 9.8.4 | Ocular symptoms | 27 |
| 9.8.5 | Visual acuity | 28 |
| 9.8.6 | Slit lamp examination | 28 |
| 9.8.7 | Corneal fluorescein staining and fundus ophthalmoscopy | 28 |
| 9.8.8 | Intraocular pressure | 28 |
| 9.9 | Analysis datasets | 28 |
| 10 | REFERENCES | 29 |
| 11 | APPENDICES | 30 |





#### ABBREVIATIONS

AE Adverse Event

CA Competent Authority

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval
CPL Clinical Project Leader
CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organisation

CSP Clinical Study Protocol
CSR Clinical Study Report
CV Coefficient of Variation
EC Ethics Committee
ETV Early Termination Visit

FDA Food and Drug Administration

FSFV First Subject First Visit GCP Good Clinical Practice

ICH International Conference on Harmonisation

IGA Investigator Global Assessment
IMP Investigational Medicinal Product

IP Investigational Product LSLV Last Subject Last Visit

MedDRA Medical Dictionary for Regulatory Activities

NA Not Applicable
NC Not calculated
OTC Over The Counter
PT Preferred Term

PTAE Pre-Treatment Adverse Event

SAE Serious Adverse Event SD Standard Deviation SOC System Organ Class

SOP Standard Operating Procedure SDTM Study Data Tabulation Model

TEAE Treatment-Emergent Adverse Event
USDA United States Department of Agriculture

WHODDE World Health Organisation Drug Dictionary Enhanced



#### 1 INTRODUCTION

Statistical analysis will be performed by the CROSS Research Biometry Unit. The end-points and methods of analysis specified in this SAP are consistent with ICH E6 (R2) and E9 guidelines (1, 2). The SAP has been compiled by the CRO Biometry Unit on the basis of the final version 1.0 of the clinical study protocol and its amendment (3, 4), reviewed by the Sponsor and finalized before the database lock and the treatment unblinding.

# 1.1 Changes with respect to the study protocol and its amendment(s)

The following changes were introduced in the SAP with respect to the study protocol and its amendment (3, 4):

- Body weight will not be treated as a safety assessment (§9.2 of study protocol), because collected only at screening
- Changes from baseline for values or scores for Corneal fluorescein staining and fundus ophthalmoscopy parameters will not be evaluated



#### 2 STUDY/INVESTIGATON OBJECTIVES

The objective of the study is to evaluate the efficacy, safety and local tolerability of Chloroprocaine 3% ophthalmic gel as compared to matching placebo in healthy subjects.

#### 2.1 Primary end-point

Proportion of subjects gaining full conjunctival anesthesia of the ocular surface, evaluated by conjunctiva pinching (0.3-mm forceps), 5 minutes after administration of Chloroprocaine 3% ophthalmic gel, in comparison to placebo - only study eye (right eye).

#### 2.2 Secondary end-points

- Time to anesthesia, evaluated by conjunctiva pinching (0.3-mm forceps) only study eye (right eye)
- Duration of anesthesia, evaluated by conjunctiva pinching (0.3-mm forceps) only study eye (right eye)
- Visual acuity both eyes
- Ocular symptoms (burning, stinging, itching, foreign body sensation) evaluated using a 0-100 mm VAS both eyes
- Objective ocular signs (Conjunctival redness, anterior chamber flare, conjunctival chemosis, eyelid swelling) by Slit lamp examination both eyes
- Corneal fluorescein staining by slit lamp examination both eyes
- Intraocular pressure (IOP) both eyes
- Fundus ophthalmoscopy (vitreous, macula, retina and optic nerve head) with the slit lamp both eyes
- Treatment-emergent adverse events (TEAEs), assessed throughout the study
- Vital signs (blood pressure and heart rate)



#### 3 INVESTIGATIONAL PLAN

#### 3.1 Overall study design

This is a phase I/II, single dose, randomised, placebo-controlled, parallel-group, double-masked, efficacy, safety and local tolerability study.

#### 3.2 Discussion of design

This study was performed as part of a clinical development program for Chloroprocaine 3% ophthalmic gel, following scientific advice obtained from the FDA in Sept. 2019.

The study enrolled a total of 105 healthy men and women. According to the study design, initially safety and local tolerability was evaluated on the data collected for the first 20 randomised subjects (16 treated with the active product and 4 with placebo). For these subjects, no efficacy evaluation was carried out. Because safety and local tolerability were confirmed after the first enrolled subjects, the study continued with the following 85 men and women (68 treated with the active product and 17 with placebo) on which treatment efficacy as well as safety was assessed.

Each randomised subject was allocated to a treatment group according to a computer generated randomisation list and a 4: 1 ratio for active treatment vs. placebo. The study was double-masked and the two investigational products were indistinguishable.

See the clinical study protocol and its amendment (3, 4) for further details.



#### 4 STUDY POPULATION

#### 4.1 Target population

Healthy male and female subjects, aged 18-55 years inclusive.

#### 4.2 Inclusion criteria

To be enrolled in this study, subjects had to fulfil all these criteria:

- 1. Informed consent: signed written informed consent before inclusion in the study
- 2. Sex and age: Healthy men and women, 18 55 years inclusive
- 3. Body Mass Index: 18.5-30 kg/m<sup>2</sup> inclusive
- 4. *Vital signs*: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest in the sitting position
- 5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study
- 6. Contraception and fertility: women of child-bearing potential must be using at least one of the following reliable methods of contraception:
  - a. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit;
  - b. A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
  - c. A male sexual partner who agrees to use a male condom with spermicide
  - d. A sterile sexual partner

Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. For all women, urine pregnancy test result must be negative at screening.

#### 4.3 Exclusion criteria

Subjects meeting any of these criteria could not be enrolled in the study:

- 1. Physical findings: Clinically significant abnormal physical findings which could interfere with the objectives of the study
- 2. Visual acuity: Best corrected visual acuity < 1/10
- 3. Concomitant medications: Medications, including over the counter medications and herbal remedies, systemic opioids and morphine drugs, topical ocular products with anaesthetic action, systemic analgesic drugs, for 2 weeks before study screening
- 4. Ophthalmic diseases: Clinically significant ocular disease; eye movement disorder (i.e. nystagmus); dacryocystitis and all others pathologies of tears drainage system; corneal, epithelial, stromal or endothelial, residual or evolutionary disease (including corneal ulceration and superficial punctuate keratitis); history of inflammatory ocular disease (iritis, uveitis, herpetic keratitis), history of ocular traumatism, infection or inflammation



- within the last 3 months or history of any other ocular disease that may affect the outcome of the study or the subject's safety
- 5. Ophthalmic surgery: History of ophthalmic surgical complications (e.g. cystoid macular oedema) in the last 6 months
- 6. *Diseases*: Significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine, psychiatric or neurological diseases or surgeries that may interfere with the aim of the study
- 7. Allergy: Ascertained or presumptive hypersensitivity to the active principle and/or ingredients of investigational products; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study
- 8. *Investigative drug studies*: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
- 9. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to the USDA Dietary Guidelines 2015-2020], caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥10 cigarettes/day)
- 10. Alcohol test: positive alcohol breath test at Day 1
- 11. Pregnancy (women only): positive or missing pregnancy test at screening, pregnant or lactating women

#### 4.3.1 Not allowed treatments

Any medications, including over the counter (OTC) and herbal remedies, in particular systemic opioids and morphine drugs, topical ocular products with anaesthetic action and systemic analgesic drugs, were NOT allowed for 2 weeks before the start of the study and during the whole study duration. Paracetamol was allowed as therapeutic counter-measure for adverse events (AEs) according to the Investigator's opinion. Hormonal contraceptives were allowed.

The intake of any other medication will be reported as a protocol deviation. However, it lead to subject's discontinuation from the study only if the Investigator, together with the Sponsor, considers it could affect the study assessments or outcome.



#### 5 STUDY SCHEDULE

The schedule of the study is summarised at page 5.

#### 5.1 Study visits and procedures

Each study subject underwent 4 visits.

The study protocol foresees 1 period for each subject. Maximum study duration was 29 days, screening visit and follow-up included. A written informed consent was obtained before any study assessment or procedure.

The first subject first visit (FSFV) is defined as the 1<sup>st</sup> visit performed at the clinical centre by the 1<sup>st</sup> screened subject. The last subject last visit (LSLV) is defined as the last visit performed at the clinical centre by the last subject, i.e. the last visit foreseen by the study protocol, independently of the fact that the subject is a completer or a withdrawn subject.

The following phases, visits and procedures were performed:

- Screening phase
  - Screening visit 1: day -21 / day -1
- Interventional phase
  - Visit 2: day 1
- Final phase
  - Visit 3: day 2: Telephone call
  - Visit 4: day  $7 \pm 1$  or at early discontinuation: follow-up/early termination visit (ETV).

The schedule of the study procedures and assessments is presented below:



# **Schedule:**

| | Day | Procedures/Assessments |
|---|---|---|
| | Day | Explanation to the subject of study aims, procedures and possible risks |
| | | <ul> <li>Informed consent signature</li> </ul> |
| | | <ul> <li>Screening number (as S001, S002, etc.)</li> </ul> |
| | | > Demographic data |
| | | <ul> <li>Ocular medical and surgical history</li> </ul> |
| | | <ul> <li>Other medical and surgical history</li> </ul> |
| 1 | | <ul> <li>Previous and concomitant medications</li> </ul> |
| Screening – Visit 1 | | <ul> <li>Physical examination (including ocular examination, body weight, height)</li> </ul> |
| ·Vi | | > Vital signs (blood pressure and heart rate) check |
| 5.0 | Day -21 / | > Urine pregnancy test for women |
| nin | Day -1 | Adverse event (AE) monitoring |
| ree | , | Coular symptoms (0-100 mm VAS) - all subjects - both eyes |
| Sci | | ➤ Visual acuity (EDTRS) – both eyes |
| | | > Slit lamp examination (SLE; Conjunctival redness, anterior chamber flare, conjunctival |
| | | chemosis, eyelid swelling) - all subjects - both eyes |
| | | Corneal fluorescein staining with SLE - all subjects - both eyes |
| | | > Intraocular pressure measurement - all subjects - both eyes |
| | | Fundus ophthalmoscopy (with slit lamp) - all subjects - both eyes |
| | | > Inclusion/exclusion criteria evaluation |
| | | > Eligibility evaluation |
| | | ➤ Alcohol test |
| | | > Inclusion/exclusion criteria evaluation |
| | | > Subject eligibility confirmation |
| | | > Enrolment and randomisation |
| | | Vital signs (blood pressure, heart rate) check - pre-dose - all subjects |
| | | Coular symptoms (0-100 mm VAS) - pre-dose - all subjects - both eyes |
| | | > Slit lamp examination (SLE; Conjunctival redness, anterior chamber flare, conjunctival |
| | | chemosis, eyelid swelling) - pre-dose - all subjects - both eyes |
| Visit 2 | | Instillation of the investigational product (right eye only) |
| Vis | Day 1 | Assessment of conjunctival anaesthesia by conjunctival pinching (0.3 mm forceps) at |
| | | the pre-specified post-dose assessment times - efficacy evaluation subjects only - study eye only (right eye) |
| | | <ul> <li>Ocular symptoms (0-100 mm VAS) - at the end of the study day - all subjects - both</li> </ul> |
| | | eyes |
| | | <ul> <li>Vital signs (blood pressure, heart rate) check - at the end of the study day - all subjects</li> </ul> |
| | | > Slit lamp examination - at the end of the study day (SLE; Conjunctival redness, |
| | | anterior chamber flare, conjunctival chemosis, eyelid swelling) - all subjects - both |
| | | eyes |
| | | AE and concomitant medications (throughout the study day) |
| 3 | Day 2 - | |
| Visit 3 | Phone | > AE and concomitant medications check |
| > | call | |
| | ı | |



# **Schedule, continued:**

| | Day | Procedures/Assessments |
|---|---|---|
| | | ➤ AE and concomitant medications |
| | | ➤ Vital signs (blood pressure, heart rate) check |
| | | > Physical examination |
| | | Coular symptoms (0-100 mm VAS) - both eyes |
| it 4 | Day $7 \pm 1$ | ➤ Visual acuity (EDTRS) – both eyes |
| Visit | Follow up | Slit lamp examination (SLE; Conjunctival redness, anterior chamber flare, conjunctival chemosis, eyelid swelling) - both eyes |
| | | Corneal fluorescein staining (with SLE) - both eyes |
| | | > Intraocular pressure measurement - both eyes |
| | | Fundus ophthalmoscopy (with slit lamp) - all subjects - both eyes |

# 5.2 Diet and lifestyle

Not applicable.



# 6 STUDY SUBJECT IDENTIFICATION METHOD AND TREATMENT ASSIGNMENT METHOD

# 6.1 Unique subject identifier

All the subjects who signed the informed consent form for the present study were coded with "unique subject identifiers" when data were extracted from the study database into the domains of the CDISC SDTM model. The unique subject identifier consists of the Sponsor study code (i.e. CHL.3-01-2020), the 3-digit site number (i.e. 001), the 4-digit screening number (e.g. S001, S002, etc.) and, if applicable, the 3-digit subject randomisation number (e.g. 001, 002, etc.). Study code, site number, screening number and subject randomisation number are separated by slashes ("/").

# 6.2 Subject identifier for the study

The last 8 digits of the unique subject identifier (enrolled subjects), corresponding to the subject screening and subject randomisation numbers separated by a slash, or the last 4 digits of the unique subject identifier (not enrolled subjects), corresponding to the subject screening number, will appear as subject identifier in the individual listings and figures of the clinical study report.

#### 6.3 Randomisation

The randomisation list was computer-generated by the Biometry Unit of the Clinical Contract Research Organization (CRO), using the PLAN procedure of the SAS® version 9.3 (TS1M1) (5) according to the following specification:

• Allocation ratio: 4:1

Randomisation method: SimpleStratification factors: None

The randomisation list will be attached to the final clinical study report.

#### 6.4 Treatment allocation

Subjects were assigned to one of the two treatment groups (Choroprocaine/placebo) in a 4:1 ratio according to the randomisation list. A randomisation number was given to the subjects on study day 1 in chronological order, after eligibility confirmation.

#### 6.5 Blinding

The study was carried out in a double-masked (double-blind) fashion, therefore the Investigator/deputy administering the investigational products, the ophthalmologists performing the measurements as well as the study participants didn't know the allocated product.

Three (3) copies of the randomisation list were generated and sealed in individual envelopes:

> one copy was sent to the manufacturer for the preparation of the individual treatment boxes



- > one copy is kept at the CRO Quality Assurance Unit
- > one copy is stored in the statistical study file

Neither the members of the clinical unit nor the CPL or the CRA/monitor will have access to the randomisation code.

The CRO will open the envelope containing the randomisation list only when data-entry is complete and decisions to be made in blinding, before data analysis, are final.

The CRO will notify breaking of the randomisation list to the Sponsor.

# **6.5.1** Emergency code and unblinding procedures

Unblinding of the code for specific subjects, if applicable, was fully documented in the source documents and in the clinical study report.

#### 6.5.2 Emergency individual envelopes

Inside the envelope, the randomisation code must be clearly indicated, reporting the allocated treatment.

The true randomisation code is filed in the Investigator's study file in a sealed envelope for each subject, with the key for its identification. Copies of the emergency individual envelopes were sent to the pharmacovigilance representative and to the Sponsor representative (if not coinciding).

Breaking of an individual randomisation code, by the Investigator during the study, was allowed only when knowledge of the code by the Investigator was essential for the subject's health. In these cases, the Investigator opens only the envelope related to the concerned subject. Individual code breaking is clearly reported in the subject-related CRF and the envelope itself; the latter is sealed again.

In any case, the CRA/monitor must be informed within 24 h from code breaking.

The date and the reason for breaking the code must be recorded in the CRF and on the envelope. All envelope sets containing the randomisation code of each subject must be kept closed even after database lock. At the end of the study, all envelope sets will be sent to the Sponsor.

No breaking of individual randomisation codes occurred during the study.



#### 7 STUDY EVALUATION PARAMETERS

#### 7.1 Study variables

#### 7.1.1 Primary variables

• Conjunctival anaesthesia evaluation by conjunctival pinching (with 0.3 mm forceps) at 5 min post-dose - only study eye (right eye).

# 7.1.2 Secondary variables

- Conjunctival anaesthesia evaluation by conjunctival pinching (with 0.3 mm forceps) at the pre-specified assessment time-points (see below) only study eye (right eye)
- Ocular symptoms (burning, stinging, itching, foreign body sensation) using a 0-100 mm VAS- both eyes
- Visual acuity (EDTRS chart) both eyes
- Objective ocular signs (Conjunctival redness, anterior chamber flare, conjunctival chemosis, eyelid swelling) by SLE- both eyes
- Corneal fluorescein staining by SLE- both eyes
- Intraocular pressure (IOP) both eyes
- Fundus ophthalmoscopy (vitreous, macula, retina and optic nerve head) with the slit lamp-both eyes
- Treatment-emergent adverse events (TEAEs), assessed throughout the study
- Vital signs (blood pressure and heart rate).

#### 7.2 Safety assessments

Safety and general tolerability of the investigational products will be based on TEAEs, ocular symptoms (0-100 mm VAS), physical examinations including body weight, vital signs, visual acuity, SLE, corneal fluorescein staining, fundus ophthalmoscopy and IOP results.




#### 8 DATA MONITORING COMMITTEE AND BLIND REVIEW MEETING

#### 8.1 Composition of data monitoring committee

No data monitoring committee was established for this study.

# 8.2 Purpose and scope of the blind review meeting

According to ICH and EMA guidelines (1, 2), the main objectives of the blind review meeting are:

- definition of analysis sets
- review of the protocol deviations
- review of the current version of the SAP
- detection and discussion of any other relevant data issue, which may affect the analysis

Analysis sets definition, protocol deviations and data issues have to be reviewed on a case-by-case basis by the study team, before database lock.




#### 9 STATISTICAL METHOD

The statistical analysis of demographic, baseline and background characteristics, efficacy, safety and tolerability data will be performed using SAS® version 9.3 (TS1M1) (5) or higher (the actual versions will be stated in the final report).

The data documented in this study and the parameters measured will be evaluated and compared using classic descriptive statistics, i.e. arithmetic mean, SD, CV (%), minimum, median and maximum values for quantitative variables and frequencies for qualitative variables

Not available data will be evaluated as "missing values".

#### 9.1 Tables, listings and figures layout

Tables, listings and figures will be provided according to the following settings:

- Background: White
- Foreground: Black
- Font face: Times
- Font style: Roman
- Font size: 10 pt
- Font weight: Medium (data, footers and notes), Bold (titles and headers)
- Font width: Normal
- Layout: Landscape
- Top Margin: 2.5 cm
- Bottom Margin: 2.5 cm
- Left Margin: 0.8 cm
- Right Margin: 0.8 cm
- Test label: Chloroprocaine 3% ocular gel
- Control label: Placebo
- Date format: ddMMMyyyy
- Means, standard deviations, percent coefficient of variations, medians, lower confidence limits and upper confidence limits will be rounded to one digit more than the original data
- Minima and maxima will keep the same number of decimal digits as the source values
- p-values will be rounded to the fourth decimal digit and will be flagged by an asterisk (\*) in case of statistical significance (i.e. p-value < 0.05 or, in case of centre by treatment interaction, p-value < 0.10)
- p-values lower than 0.0001 will be reported as "<.0001 \*".

The data and results of Chloroprocaine 3% ocular gel will be presented before the data and results of Placebo in all listings and tables.

#### 9.2 Analysis sets

#### 9.2.1 Definitions



A subject will be defined as <u>screened</u> after the signature of the informed consent, regardless of the completion of all the screening procedures.

A subject will be defined as eligible if he/she meets all the inclusion/exclusion criteria. Otherwise he/she will be defined as a screen failure.

A subject will be defined as <u>enrolled</u> in the study if he/she is included in the interventional phase of the study. The enrolment will be performed through randomised allocation to a treatment arm

An eligible but not enrolled subject will be defined as a reserve.

A subject will be defined as <u>randomised</u> in the study when he/she is assigned to a randomised treatment arm.

The following data sets will be used for the analysis:

- *Enrolled Set*: all enrolled subjects. This analysis set will be used for demographic, baseline and background characteristics
- Full Analysis Set (FAS): all randomised subjects, who receive the dose of the investigational product and have at least one post randomisation assessment of the primary efficacy data. This analysis set will be used for the primary efficacy analysis
- Per Protocol Set (PP): all randomised subjects who fulfil the study protocol requirements in terms of investigational product intake and collection of primary efficacy data and with no major deviations that may affect study results. This analysis set will be used for sensitivity analyses
- Safety Set: all subjects who receive at least one dose (drop) of the investigational product. This analysis set will be used for the safety analyses

Each subject will be coded by the CRO Biometry Unit as valid or not valid for the Enrolled Set, Full Analysis Set, Per Protocol Set and Safety Set before database lock and treatment unblinding. Subjects will be evaluated according to the treatment they actually received (Enrolled Set, Full Analysis Set, Per Protocol Set and Safety Set).

#### 9.2.2 Reasons for exclusion from the Full Analysis Set

According to ICH E9 guideline (2), the reasons for exclusion of subjects from the Full Analysis Set are the following:

- failure to take the investigational product
- lack of any primary efficacy data post enrolment
- failure to satisfy major inclusion/exclusion criteria (eligibility deviations). Subjects who fail to satisfy an inclusion/exclusion criterion may be excluded from the analysis without the possibility of introducing bias only under the following circumstances:
  - the inclusion/exclusion criterion was measured prior to enrolment
  - the detection of the relevant eligibility deviations is completely objective
  - all subjects receive equal scrutiny for eligibility deviations (blind review)



all detected deviations of the particular inclusion/exclusion criterion are excluded

#### 9.2.3 Reasons for exclusion from the Per Protocol Set

Reasons for exclusion of subjects from the Per Protocol Set include (but are not limited to) the following:

- lack of compliance to the investigational product
- exposure to an investigational product different from the one assigned to the subject
- missing primary efficacy data
- failure to satisfy any inclusion/exclusion criteria (eligibility deviations)
- intake of prohibited medications

The precise reasons for excluding subjects from the Per Protocol Set will be fully defined and documented during the blind review meeting before breaking the blind.

#### 9.2.4 Reasons for exclusion from the Safety Set

Reason for exclusion of subjects from the Safety Set is the following:

• failure to take at least one dose (drop) of the investigational product

#### 9.3 Sample size and power considerations

A total of 105 healthy men and women will be included in the study. Active vs. placebo treatment will have a 4:1 ratio.

Initially, local tolerability and safety will be evaluated on the first 20 enrolled subjects (16 treated with chloroprocaine 3% ocular gel and 4 with placebo).

After the first 20 subjects have completed the study, local tolerability and safety data will be evaluated and if treatment safety is confirmed, efficacy, beside local tolerability and safety, will be assessed on the 85 subsequent subjects (68 active gel and 17 with placebo).

Sample size for the efficacy evaluation was formally calculated as follows:

Sample size per group was calculated by comparing two independent proportions (experimental and placebo success rate) with a two-sided alpha=0.05 and a power of 0.95. This is based on the assumption, that the experimental success rate is 80% and the vehicle success rate is 30%, taking a dropout rate of 20% into account. For sample size estimation, NQuery (Version 4.0) was used implementing formulas described in Chow et al (2008) (7).



# 9.4 Demographic, baseline and background characteristics

Demographic, baseline and background characteristics will be reported for all the enrolled subjects and analyses will be performed according to the treatment they actually received (Enrolled Set, Full Analysis Set, Per Protocol Set, Safety Set).

# 9.4.1 Subjects' disposition

The disposition of all subjects enrolled in the study will be listed (Listing 16.2.4.1) and summarised (Table 14.1.1.1). The number and proportion of subjects enrolled, randomised, treated and completing the study, the number and proportion of withdrawals and the reasons for withdrawal will be presented.

#### 9.4.2 Analysis sets

The subjects included in each analysis sets will be listed (Listing 16.2.4.2) and summarised by treatment group (Table 14.1.1.2).

#### 9.4.3 Subjects excluded from efficacy and/or safety analysis

All subjects excluded from the efficacy and/or safety analysis will be listed (Listing 16.2.3.1) and the reasons for exclusion will be reported.

#### 9.4.4 Discontinued subjects

All subjects who discontinued the clinical trial (if any) will be listed (Listing 16.2.1.1). Last IP administered before discontinuation, gender, age, last visit performed before discontinuation, time elapsed from last IP administration (days), date of premature discontinuation and primary reason for subject premature discontinuation will be reported.

#### 9.4.5 Protocol deviations

All the protocol deviations reported during the clinical trial will be listed (Listing 16.2.2.1) and summarised (Table 14.1.1.5). The number and proportion of subjects for each deviation will be reported.

#### 9.4.6 Treatment mismatch

All subjects with actual treatment arm different from assigned treatment arm will be listed (Listing 16.2.2.2).

#### 9.4.7 **Demography**

Demographic data will be listed (Listing 16.2.4.3) and summarised (Table 14.1.1.3). The number and proportion of subjects in each category for categorical variables (e.g. sex, race) and descriptive statistics (mean, SD, CV%, minimum, median and maximum) for continuous variables (e.g. age, weight) will be presented.



#### 9.4.8 Inclusion/exclusion criteria not met

All the unmet inclusion/exclusion criteria will be listed (Listing 16.2.4.4) and summarised (Table 14.1.1.4).

#### 9.4.9 Medical and surgical history

All the diseases of ocular history and medical history, ocular surgery and other surgeries of all subjects enrolled in the study will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 23.1 or higher, and listed (Listing 16.2.10.1).

#### 9.4.10 Prior and concomitant medication

All prior and concomitant medications will be coded using the World Health Organization Drug Dictionary Enhanced (WHODDE), version September 2020 or higher, and listed (Listing 16.2.10.3).

#### 9.4.11 Subjects' study visits

The dates of all subjects study visits will be listed (Listing 16.2.10.4).

#### 9.4.12 Fertility status and contraceptive method

The fertility status and the contraceptive method used by the subjects will be listed (Listing 16.2.10.5).

#### 9.4.13 Alcohol breath test and pregnancy test

The date/time and the result of alcohol breath test and pregnancy test will be listed (Listing 16.2.8.1).

#### 9.5 IMP administration

The date and time of all IMP administrations will be listed (Listing 16.2.5.1).

#### 9.6 Interim analyses

No interim analysis was planned for the study.

#### 9.7 Efficacy analysis

#### 9.7.1 Primary efficacy analysis

The primary efficacy analysis will be performed on the subjects included into the Full Analysis Set.

Subjects will be analysed according to the treatment they actually received.



Primary end-point is defined as the proportion of subjects gaining full anesthesia of the ocular surface 5 minutes after administration of the investigational product for the 2 treatment arms (cornea pinching assessment).

The date/time and the results of cornea pinching assessments will be listed (Listing 16.2.6.1)

The result of the anesthesia will be coded as success/failure, listed by subject (Listing 16.2.6.2) and summarised (Table 14.2.1.1) overall and by treatment group using contingency tables. Resulting proportions will be presented together with 95% confidence interval. The 2 groups (active and placebo) will be compared using Pearson's  $\chi^2$  test. The null hypothesis of equal success between the 2 treatment arms at the  $\alpha$ =0.05 level will be rejected if:

$$\left| \frac{\widehat{p_1} - \widehat{p_2}}{\sqrt{\frac{\widehat{p_1}(1 - \widehat{p_1})}{n_1} + \frac{\widehat{p_2}(1 - \widehat{p_2})}{n_2}}} \right| > Z_{\alpha/2}$$

where  $p_1$  is the proportion of subjects who meet the primary endpoint in the active group, while  $p_2$  is the proportion of subjects who meet the primary endpoint in the vehicle (placebo) group.

#### 9.7.2 Sensitivity analyses

The primary efficacy analysis will be repeated in the Per Protocol Set (Table 14.2.1.2) in order to evaluate the robustness of the results obtained on the Full Analysis Set. Subjects will be analysed according to the treatment they actually received.

#### 9.7.3 Secondary efficacy analysis

The secondary efficacy analysis will be performed on the subjects included into the Full Analysis Set and in the Per Protocol Set. Subjects will be analysed according to the treatment they actually received.

Time to anesthesia and duration of anesthesia will be listed (Listing 16.2.6.2) and summarised overall and by group using descriptive statistics (mean, median, standard deviation, minimum, maximum, 95% confidence interval on the mean, and number of observations). The 2 groups (active and placebo) will be compared using non-parametric Mann-Whitney's test for continuous variables (Table 14.2.2.1, Table 14.2.2.2).

#### 9.8 Safety and tolerability analysis

The safety and tolerability analysis will be performed on the subjects included into the Safety Set

Subjects will be analysed according to the treatment they actually received.

#### 9.8.1 Adverse events



Adverse events (AEs) will be coded by System Organ Class (SOC) and Preferred Term (PT), using the Medical Dictionary for Regulatory Activities (MedDRA) version 23.1 or higher. AEs will be classified as pre-treatment AEs (PTAEs) and treatment-emergent AEs (TEAEs), according to the period of occurrence, as follows:

- PTAEs: all AEs occurring before the first dose of IMP and not worsening after the first dose of IMP
- TEAEs: all AEs occurring or worsening after the first dose of IMP

Individual PTAEs and TEAEs will be listed in subject data listings (Listing 16.2.7.2, Listing 16.2.7.1).

No summary table will be provided for PTAEs.

TEAEs will be summarised by treatment group and overall. The number and percentage of subjects with any TEAE and the number of TEAEs will be presented overall and by SOC and PT, seriousness, relationship to treatment and severity. (Table 14.3.1.1, Table 14.3.1.2, Table 14.3.1.3, Table 14.3.1.4). For TEAEs that change severity during the study (e.g. from mild to moderate or from moderate to mild), the most severe intensity will be reported in the summary tables.

Should any serious TEAE occur, the number and percentage of subjects with any serious TEAE, the number of serious TEAEs, the number and percentage of subjects with any serious TEAE related to study drug and the number of serious TEAEs related to study drug will be presented (Table 14.3.1.5, Table 14.3.1.6).

All TEAEs leading to death, serious TEAEs and TEAEs leading to discontinuation will be listed, if applicable (Table 14.3.2.1).

#### 9.8.2 Vital signs

The date/time of vital signs assessments and the values of vital signs will be listed (Listing 16.2.9.1) and summarised using descriptive statistics at screening and end of study (Table 14.3.5.2) and by treatment during the study (Table 14.3.5.3).

A table of all the abnormal vital signs' values will be presented (Table 14.3.5.1).

#### 9.8.3 Physical examination

The date of physical examination and the overall investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant) and clinically significant abnormalities (if any) will be listed (Listing 16.2.10.2).

#### 9.8.4 Ocular symptoms

The date/time of ocular symptoms assessments and the VAS scores for ocular tolerability parameters (burning, stinging, itching, foreign body sensation) and their changes from baseline will be listed (Listing 16.2.9.2) and summarised (Table 14.3.5.4) by treatment and



eye using descriptive statistics (mean, SD, CV%, minimum, median and maximum). Changes from baseline will be evaluated and compared between treatments. (Table 14.3.5.5)

#### 9.8.5 Visual acuity

The date/time of assessments and the visual acuity results will be listed (Listing 16.2.9.3) by subject and summarised (Table 14.3.5.6) for each eye by descriptive statistics.

#### 9.8.6 Slit lamp examination

The date/time of assessments and the values for Slit lamp examination (SLE) parameters and their changes from baseline will be listed (Listing 16.2.9.4) and summarised (Table 14.3.5.7) for each eye using descriptive statistics (mean, SD, CV%, minimum, median and maximum).

#### 9.8.7 Corneal fluorescein staining and fundus ophthalmoscopy

The date/time of assessments and the values or scores for Corneal fluorescein staining and Fundus ophthalmoscopy parameters will be listed (Listing 16.2.9.5, Listing 16.2.9.6) and summarised (Table 14.3.5.8, Table 14.3.5.9) for each eye by descriptive statistics.

#### 9.8.8 Intraocular pressure

The date/time of intraocular pressure assessments and the IOP values will be listed (Listing 16.2.9.7) and summarised (Table 14.3.5.10) for each eye by descriptive statistics.

#### 9.9 Analysis datasets

Analysis datasets will be created according to the version 2.1 of the ADaM model of CDISC (8).



#### 10 REFERENCES

- 1 ICH Topic E6 (R2): Good clinical practice.
- 2 ICH Topic E9: Statistical principles for clinical trials.
- 3 Study Protocol CRO-PK-20-343. A Phase I/II, randomized, placebo-controlled, double-masked, efficacy, safety and local tolerability study of Chloroprocaine 3% gel eye drops in healthy volunteers. Final version 1.0, 21FEB2020
- 4 Study Protocol CRO-PK-20-343. A Phase I/II, randomized, placebo-controlled, double-masked, efficacy, safety and local tolerability study of Chloroprocaine 3% gel eye drops in healthy volunteers. Amendment Nr. 1, Final version 1.0, 05AUG2020
- 5 SAS/STAT® User's Guide
- 6 Phoenix 1.3 User's Guide, Pharsight Corporation
- 7 Chow S-C, Shao J, Wang H. Sample size calculations in clinical research: Chapman and Hall/CRC; 2008
- 8 CDISC Analysis Data Model Version 2.1





#### 11 APPENDICES

- 1. Section 14 Tables and Figures Shells
- 2. Section 16.2 Individual Subject Data Listings Shells




Statistical analysis plan CRO-PK-20-343 Sponsor code CHL.3-01-2020 Chloroprocaine 3% ocular gel Final version 1.0, 20NOV20

#### Section 14 - Tables Shells

| Table 14.1.1.1 - Subjects' dispos | sition - Enrolled set |
|-----------------------------------|-----------------------|
|-----------------------------------|-----------------------|

- Table 14.1.1.2 Analysis sets Enrolled set
- Table 14.1.1.3 Demography Enrolled set, Safety set, Full Analysis set and Per Protocol set
- Table 14.1.1.4 Inclusion/exclusion criteria not met Enrolled set, Safety set, Full Analysis set and Per Protocol set
- Table 14.1.1.5 Protocol deviations Enrolled set, Safety set, Full Analysis set and Per Protocol set
- Table 14.2.1.1 Anesthesia proportion of success Full analysis set
- Table 14.2.1.2 Anesthesia proportion of success Per Protocol set
- Table 14.2.2.1 Anesthesia results Full Analysis set
- Table 14.2.2.2 Anesthesia results Per Protocol set
- Table 14.3.1.1 Global incidence of subjects with treatment-emergent adverse events Safety set
- Table 14.3.1.2 Subjects with treatment-emergent adverse events by system organ class and preferred term Safety set
- Table 14.3.1.3 Subjects with treatment-emergent adverse events by intensity, system organ class and preferred term Safety set
- Table 14.3.1.4 Subjects with treatment-emergent adverse events related to the IP by system organ class and preferred term Safety set
- Table 14.3.1.5 Subjects with serious treatment-emergent adverse events by system organ class and preferred term Safety set
- Table 14.3.1.6 Subjects with serious treatment-emergent adverse events related to the IP by system organ class and preferred term Safety set
- Table 14.3.2.1 Treatment-emergent adverse events leading to death, serious or leading to discontinuation Safety set
- Table 14.3.5.1 Abnormal vital signs Safety set
- Table 14.3.5.2 Descriptive statistics of vital signs at screening and end of study Safety set
- Table 14.3.5.3 Descriptive statistics of vital signs during the study Safety set
- Table 14.3.5.4 Descriptive statistics of ocular symptoms Safety set
- Table 14.3.5.5 Wilcoxon Rank Sum Test on changes from baseline in Ocular Symptoms Safety set
- Table 14.3.5.6 Descriptive statistics of visual Acuity Safety set
- Table 14.3.5.7 Descriptive statistics of slit lamp examination Safety set
- Table 14.3.5.8 Descriptive statistics of corneal fluorescein staining Safety set
- Table 14.3.5.9 Descriptive statistics of fundus ophthalmoscopy Safety set
- Table 14.3.5.10 Descriptive statistics of intraocular pressure Safety set




#### Table 14.1.1.1 - Subjects' disposition - Enrolled set

| | Overall<br>n (%) |
|--------------------------------------------|------------------|
| Enrolled | nn |
| Enrolled but not randomised <sup>1</sup> | nn (xx.x) |
| Randomised <sup>1</sup> | nn (xx.x) |
| Discontinued before treatment <sup>2</sup> | nn (xx.x) |
| Treated <sup>2</sup> | nn (xx.x) |
| Completed <sup>3</sup> | nn (xx.x) |
| Discontinued <sup>3</sup> | nn (xx.x) |
| Adverse event <sup>3</sup> | nn (xx.x) |
| Withdrawal by subject <sup>3</sup> | nn (xx.x) |
| | nn (xx.x) |

Note: The number and the proportion of subjects of each disposition event are reported

Note 1: The denominator for calculating the proportion is the number of enrolled subjects

Note 2: The denominator for calculating the proportion is the number of randomised subjects

Note 3: The denominator for calculating the proportion is the number of randomised and treated subjects

Source: Listing 16.2.4.1 - Subjects' disposition

Program: Tables\k343-ds-tbl.sas



Table 14.1.1.2 - Analysis sets - Enrolled set

| | | <b>Enrolled Set</b> | |
|---|---|---|---|
| | Chloroprocaine 3%<br>ocular gel<br>N=XX<br>n (%) | Placebo<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
| Safety Set | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Full Analysis Set | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Per Protocol Set | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the product they were assigned to

The number and the proportion of subjects included in each analysis set are reported

The denominator for calculating the proportions is the number of subjects in the enrolled set of each treatment group and overall

Source: Listing 16.2.4.2 - Analysis sets

 $Program: Tables \backslash k343\text{-}ds\text{-}tbl.sas$ 



Table 14.1.1.3 - Demography - Enrolled set, Safety set, Full Analysis set and Per Protocol set

| | | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | Full Analysis Set<br>N=XX | Per Protocol Set<br>N=XX |
|---|---|---|---|---|---|---|
| Sex | Female | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | |
| | Male | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | |
| Race | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | |
| | Asian | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | |
| | Black or African American | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | |
| | White | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | |
| | Other | n (%) | nn(xx.x) | nn (xx.x) | nn (xx.x) | |
| Age [years] | | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XX | XX | XX | XX |
| Height [cm] | | N | nn | nn | nn | nn |
| <i>8</i> 1 1 | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | xx.x | XX.X | XX.X | XX.X |
| | | CV% | XX.X | xx.x | XX.X | XX.X |
| | | Min | XX | XX | XX | XX |

Note: The number and the proportion of subjects of each sex and race are reported

The denominator for calculating the proportions is the number of subjects in each analysis set

Source: Listing 16.2.4.3 - Demography Program: Tables\k343-dm-tbl.sas



Table 14.1.1.3 - Demography - Enrolled set, Safety set, Full Analysis set and Per Protocol set

| | Statistics | Enrolled Set N=XX | Safety Set<br>N=XX | Full Analysis Set<br>N=XX | Per Protocol Set<br>N=XX |
|---|---|---|---|---|---|
| Height [cm] | Median | XX.X | XX.X | XX.X | XX.X |
| | Max | XX | XX | XX | XX |
| Weight [kg] | N | nn | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | Max | xx.x | XX.X | XX.X | XX.X |
| Body Mass Index [kg/m²] | N | nn | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | Max | XX.X | XX.X | xx.x | xx.x |

Note: The number and the proportion of subjects of each sex and race are reported

The denominator for calculating the proportions is the number of subjects in each analysis set

Source: Listing 16.2.4.3 - Demography Program: Tables\k343-dm-tbl.sas



Table 14.1.1.4 - Inclusion/exclusion criteria not met - Enrolled set, Safety set, Full Analysis set and Per Protocol set

| | Enrolled Set | Safety Set | Full Analysis Set | Per Protocol Set |
|---|---|---|---|---|
| | N=XX | N=XX | N=XX | N=XX |
| Number of subjects with any inclusion/exclusion criteria not met | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criterion 1 [Informed consent] Inclusion criterion 2 [Sex and Age] | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criterion 1 [Physical findings] Exclusion criterion 2 [Visual acuity] | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: The number and the proportion of subjects for any criterion not met are reported

The denominator for calculating the proportions is the number of subjects in each analysis set

Source: Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

 $Program: Tables \verb|\k343-ie-tbl.sas|$


Table 14.1.1.5 - Protocol deviations - Enrolled set, Safety set, Full Analysis set and Per Protocol set

| | Enrolled Set<br>N=XX | Safety Set<br>N=XX | Full Analysis Set<br>N=XX | Per Protocol Set<br>N=XX |
|---|---|---|---|---|
| Number of subjects with any protocol deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Major | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Treatment deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criteria violation | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criteria violation | nn (xx.x) | nn (xx.x) | nn(xx.x) | nn (xx.x) |
| Medication not admitted | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| <del></del> | nn (xx.x) | nn (xx.x) | nn(xx.x) | nn (xx.x) |
| Minor | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled collection time | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled assessment time | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: The number and the proportion of subjects for any protocol violation are reported

The denominator for calculating the proportions is the number of subjects in each analysis set

Source: Listing 16.2.2.1 - Protocol deviations

Program: Tables\k343-dv-tbl.sas



Table 14.2.1.1 - Anesthesia proportion of success - Full analysis set

| | | Full analysis set | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Chloroprocaine 3%<br>ocular gel<br>N=XX<br>n (%) | Placebo<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) | Chloroprocaine 3%<br>ocular gel<br>Proportion<br>of success | Placebo<br>Proportion<br>of success | Difference<br>in<br>Proportions | 95%<br>two-sided<br>Confidence<br>Interval | p value<br>Chi-square<br>Test |
| Anesthesia success 1 | Y<br>N | nn (xx.x) | nn (xx.x)<br>nn (xx.x) | nn (xx.x) | | | | | |
| Chloroprocaine 3% ocular gel vs. Placebo | IN | nn (xx.x) | IIII (XX.X) | nn (xx.x) | XX.X | xx.x | xx.x | xx.x, xx.x | x.xxxx |

Note: subjects are summarised according to the product they actually received

Note 1: Anesthesia Succes is defined as full anesthesia of the ocular surface 5 minutes after administration of the investigational product

Listing 16.2.6.2 - Anesthesia results

 $Program: Tables \backslash k343\text{-eff-tbl.sas}$ 



Table 14.2.1.2 - Anesthesia proportion of success - Per Protocol set

| | | Per Protocol set | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Chloroprocaine 3%<br>ocular gel<br>N=XX<br>n (%) | Placebo<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) | Chloroprocaine 3%<br>ocular gel<br>Proportion<br>of success | Proportion | Difference<br>in<br>Proportions | 95%<br>two-sided<br>Confidence<br>Interval | p value<br>Chi-square<br>Test |
| Anesthesia success 1 | Y<br>N | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) | | | | | |
| Chloroprocaine 3% ocular gel vs. Placebo | 11 | III (AA.A) | III (AA.A) | iii (AA.A) | XX.X | xx.x | xx.x | xx.x, xx.x | x.xxxx |

Note: subjects are summarised according to the product they actually received

Note 1: Anesthesia Succes is defined as full anesthesia of the ocular surface 5 minutes after administration of the investigational product

Listing 16.2.6.2 - Anesthesia results

Program: Tables\k343-eff-tbl.sas



Table 14.2.2.1 - Anesthesia results - Full Analysis set

| | Full Analysis Set | | | | | | |
|---|---|---|---|---|---|---|---|
| | Statistics | Chloroprocaine 3%<br>ocular gel<br>N=XX | Placebo<br>N=XX | Overall<br>N=XX | Chloroprocaine 3%<br>ocular gel<br>95% CI <sup>1</sup> | Placebo<br>95% CI <sup>1</sup> | p value<br>Mann-Whitney's<br>Test |
| Time to anesthesia [min] | N | nn | nn | nn | | | |
| Time to anestnesia [mm] | Mean | XXX.X | XXX.X | XXX.X | | | |
| | SD | XXX.X | XXX.X | XXX.X | | | |
| | CV% | XXX.X | XXX.X | XXX.X | | | |
| | Min | XXX | XXX | XXX | | | |
| | Median | XXX.X | XXX.X | XXX.X | | | |
| | Max | XXX | XXX | XXX | | | |
| Time to anesthesia: Chloroprocaine 3% ocular gel vs. Placebo | | | | | xx.x, xx.x | xx.x, xx.x | x.xxxx |
| Duration of anesthesia [min] | N | nn | nn | nn | | | |
| | Mean | XXX.X | XXX.X | XXX.X | | | |
| | SD | XXX.X | XXX.X | XXX.X | | | |
| | CV% | XXX.X | XXX.X | XXX.X | | | |
| | Min | XXX | XXX | XXX | | | |
| | Median | XXX.X | XXX.X | XXX.X | | | |
| | Max | xxx | xxx | XXX | | | |
| Duration of anesthesia: Chloroprocaine 3% ocular gel vs. Placeb | o | | | | xx.x, xx.x | xx.x, xx.x | x.xxxx |

Note: Subjects are summarised according to the product they actually received

Note 1: CI is confidence interval of the mean Source: Listing 16.2.6.2 - Anesthesia results

Program: Tables\k343-eff-tbl.sas



Table 14.2.2.2 - Anesthesia results - Per Protocol set

| | | Per Protocol Set | | | | | |
|---|---|---|---|---|---|---|---|
| | Statistics | Chloroprocaine 3%<br>ocular gel<br>N=XX | Placebo<br>N=XX | Overall<br>N=XX | Chloroprocaine 3%<br>ocular gel<br>95% CI <sup>1</sup> | Placebo<br>95% CI <sup>1</sup> | p value<br>Mann-Whitney's<br>Test |
| Time to anesthesia [min] | N | nn | nn | nn | | | |
| Time to anestnesia [imiii] | Mean | XXX.X | | XXX.X | | | |
| | SD | XXX.X | XXX.X<br>XXX.X | XXX.X | | | |
| | CV% | XXX.X | XXX.X | XXX.X | | | |
| | Min | XXX | XXX | XXX | | | |
| | Median | XXX.X | XXX.X | XXX.X | | | |
| | Max | XXX | XXX | XXX | | | |
| Time to anesthesia: Chloroprocaine 3% ocular gel vs. Placebo | | | | | xx.x, xx.x | xx.x, xx.x | x.xxxx |
| Duration of anesthesia [min] | N | nn | nn | nn | | | |
| | Mean | XXX.X | XXX.X | XXX.X | | | |
| | SD | XXX.X | XXX.X | XXX.X | | | |
| | CV% | XXX.X | XXX.X | XXX.X | | | |
| | Min | XXX | XXX | XXX | | | |
| | Median | XXX.X | XXX.X | XXX.X | | | |
| | Max | XXX | xxx | XXX | | | |
| Duration of anesthesia: Chloroprocaine 3% ocular gel vs. Placeb | o | | | | XX.X, XX.X | xx.x, xx.x | x.xxxx |

Note: Subjects are summarised according to the product they actually received

Note 1: CI is confidence interval of the mean Source: Listing 16.2.6.2 - Anesthesia results

Program: Tables\k343-eff-tbl.sas



Table 14.3.1.1 - Global incidence of subjects with treatment-emergent adverse events - Safety set

| | Chloroprocaine 3%<br>ocular gel<br>N=XX<br>n (%) [n AE] | Safety Set Placebo N=XX n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
|---|---|---|---|
| Treatment-emergent Adverse Events | nn(xx.x)[kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |
| Relationship Related | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| Not related | nn(xx.x)[kk] $nn(xx.x)[kk]$ | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Intensity Mild Moderate Severe | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| Leading to discontinuation | nn (xx.x) [kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |

Note:Subjects are summarised according to the product they actually received

Subjects are summarised according to the each level of relationship and intensity reported in each treatment group and overall

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k343-ae-01-tbl.sas



Table 14.3.1.1 - Global incidence of subjects with treatment-emergent adverse events - Safety set

| | Chloroprocaine 3%<br>ocular gel<br>N=XX<br>n (%) [n AE] | Safety Set Placebo N=XX n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
|---|---|---|---|
| Serious Treatment-emergent Adverse Events | nn(xx.x)[kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |
| Relationship Related | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| Not related | nn (xx.x) [kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Intensity Mild Moderate Severe | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| Leading to discontinuation | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |

Note:Subjects are summarised according to the product they actually received

Subjects are summarised according to the each level of relationship and intensity reported in each treatment group and overall

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k343-ae-01-tbl.sas



Table 14.3.1.2 - Subjects with treatment-emergent adverse events by system organ class and preferred term - Safety set

| | Safety Set | | |
|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Chloroprocaine 3%<br>ocular gel<br>N=XX<br>n (%) [n AE] | Placebo<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Treatment-emergent Adverse Events | nn(xx.x)[kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |
| Headache | nn(xx.x)[kk] $nn(xx.x)[kk]$ | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| Gastrointestinal disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Abdominal pain upper Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version xx.x

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k343-ae-02-tbl.sas



Table 14.3.1.3 - Subjects with treatment-emergent adverse events by intensity, system organ class and preferred term - Safety set

| | Chloroprocaine 3% ocular gel N=NN Safety Set Placebo N=NN N=NN | | | | | Overall<br>N=NN | | | |
|---|---|---|---|---|---|---|---|---|---|
| System Organ Class <sup>1</sup><br>Preferred Term <sup>1</sup> | Mild<br>n (%) [n AE] | Moderate<br>n (%) [n AE] | Severe<br>n (%) [n AE] | Mild<br>n (%) [n AE] | Moderate<br>n (%) [n AE] | Severe<br>n (%) [n AE] | Mild<br>n (%) [n AE] | Moderate<br>n (%) [n AE] | Severe<br>n (%) [n AE] |
| Treatment-emergent Adverse Events | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Nervous system disorders | nn(x.x)[kk] | nn(x.x)[kk] | $nn\left( x.x\right) \left[ kk\right]$ | nn(x.x)[kk] | $nn\left( x.x\right) \left[ kk\right]$ | $nn\left( x.x\right) \left[ kk\right]$ | nn(x.x)[kk] | $nn\left( x.x\right) \left[ kk\right]$ | nn(x.x)[kk] |
| Headache | ( ) [ ] | nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk] | nn(x.x)[kk] $nn(x.x)[kk]$ | nn(x.x)[kk] $nn(x.x)[kk]$ | nn(x.x)[kk] $nn(x.x)[kk]$ | nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk] |
| Gastrointestinal disorders | nn(x.x)[kk] | nn(x.x)[kk] | $nn\left( x.x\right) \left[ kk\right]$ | $nn\left( x.x\right) \left[ kk\right]$ | $nn\left( x.x\right) \left[ kk\right]$ | $nn\left( x.x\right) \left[ kk\right]$ | $nn\left( x.x\right) \left[ kk\right]$ | $nn\left( x.x\right) \left[ kk\right]$ | nn(x.x)[kk] |
| Abdominal pain upper<br>Diarrhoea<br> | nn(x.x)[kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version xx.x

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k343-ae-02-tbl.sas



Table 14.3.1.4 - Subjects with treatment-emergent adverse events related to the IP by system organ class and preferred term - Safety set

| | Safety Set | | |
|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Chloroprocaine 3%<br>ocular gel<br>N=XX<br>n (%) [n AE] | Placebo<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Treatment-emergent Adverse Events related to the IP | nn(xx.x)[kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |
| Headache | nn(xx.x)[kk] $nn(xx.x)[kk]$ | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| Gastrointestinal disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Abdominal pain upper<br>Diarrhoea<br> | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any related adverse event and the number of related adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version xx.x

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k343-ae-02-tbl.sas



Table 14.3.1.5 - Subjects with serious treatment-emergent adverse events by system organ class and preferred term - Safety set

| | Safety Set | | |
|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Chloroprocaine 3%<br>ocular gel<br>N=XX<br>n (%) [n AE] | Placebo<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Serious Treatment-emergent Adverse Events | nn (xx.x) [kk] | nn (xx.x) [kk] | nn(xx.x)[kk] |
| Nervous system disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Headache | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| Gastrointestinal disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Abdominal pain upper Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any serious adverse event and the number of serious adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version xx.x

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k343-ae-02-tbl.sas



Table 14.3.1.6 - Subjects with serious treatment-emergent adverse events related to the IP by system organ class and preferred term - Safety set

| | | Safety Set | |
|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Chloroprocaine 3%<br>ocular gel<br>N=XX<br>n (%) [n AE] | Placebo<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Serious Treatment-emergent Adverse Events related to the IP | nn(xx.x)[kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Nervous system disorders | nn (xx.x) [kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Headache | nn(xx.x)[kk] $nn(xx.x)[kk]$ | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| Gastrointestinal disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Abdominal pain upper Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br>nn (xx.x) [kk] |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any serious related adverse event and the number of serious related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version xx.x

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k343-ae-02-tbl.sas



#### Table 14.3.2.1 - Treatment-emergent adverse events leading to death, serious or leading to discontinuation - Safety set

### Investigational Product: Chloroprocaine 3% ocular gel

| Subject | Adverse | Follow | | |
|---|---|---|---|---|
| ID | Event | Up | | |
| | ID | ID | | |
| S001/001 | 1 | | Description: | Headache |
| | | | Body Area Affected: | Head |
| | | | Preferred Term <sup>1</sup> : | Headache |
| | | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | | Acknowledgment Date/Time (Day) | ddMMMyyyy hh:mm (j) |
| | | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | | Duration: | xx h xx min |
| | | | Has the Adverse Event Started After the Administration of the Study Drug? | Y |
| | | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | | Time Elapsed form Last Study Drug intake before AE: | xx h xx min |
| | | | Reasonable Possibility of a Causal Relationship with the Study Drug? | Y |
| | | | Other Causal Relationship: | |
| | | | Severity: | Mild |
| | | | Pattern: | Continuous |
| | | | Serious Adverse Event? / Seriousness criteria: | N / |
| | | | Action taken with Study Drug: | Dose not changed |
| | | | Concomitant Therapy? | Y |
| | | | Caused Study Discontinuation? | N |
| | | | Other Action Taken: | <del></del> |
| | | | Outcome: | Recovered/Resolved |
| | | | Comments: | <del></del> |
| | | ••• | | |

Note: Subjects are listed according to the product they actually received

Note 1: MedDRA version xx.x.

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k343-ae-03-tbl.sas



#### Table 14.3.2.1 - Treatment-emergent adverse events leading to death, serious or leading to discontinuation - Safety set

### **Investigational Product: Placebo**

| Subject | Adverse | Follow | | |
|---|---|---|---|---|
| ID | Event | Up | | |
| | ID | ID | | |
| S001/001 | 2 | | Description: | Headache |
| | | | Body Area Affected: | Head |
| | | | Preferred Term <sup>1</sup> : | Headache |
| | | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | | Acknowledgment Date/Time (Day) | ddMMMyyyy hh:mm (j) |
| | | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | | Duration: | xx h xx min |
| | | | Has the Adverse Event Started After the Administration of the Study Drug? | Y |
| | | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | | Time Elapsed form Last Study Drug intake before AE: | xx h xx min |
| | | | Reasonable Possibility of a Causal Relationship with the Study Drug? | Y |
| | | | Other Causal Relationship: | <del></del> |
| | | | Severity: | Mild |
| | | | Pattern: | Continuous |
| | | | Serious Adverse Event? / Seriousness criteria: | N / |
| | | | Action taken with Study Drug: | Dose not changed |
| | | | Concomitant Therapy? | Y |
| | | | Caused Study Discontinuation? | N |
| | | | Other Action Taken: | |
| | | | Outcome: | Recovered/Resolved |
| | | | Comments: | |
| ••• | | ••• | | |

Note: Subjects are listed according to the product they actually received

Note 1: MedDRA version xx.x.

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k343-ae-03-tbl.sas



# Table 14.3.5.1 - Abnormal vital signs - Safety set

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| | ••• | <b></b> | <b></b> | ••• | ••• | ••• |

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Source: Listing 16.2.9.1 - Vital signs Program: Tables\k343-vs-tbl.sas



Table 14.3.5.2 - Descriptive statistics of vital signs at screening and end of study - Safety set

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | Screening | N | nn |
| 5,50000 51000 11 <b>0</b> 00010 [5] | Servening | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Systolic Blood Pressure [mmHg] | End of Study | N | nn |
| Systeme Brood Pressure [mm115] | End of Study | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Diastolic Blood Pressure [mmHg] | Screening | N | nn |
| | <i>g</i> | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |

Note: End of Study = Visit 4 - Follow-up or early termination visit

Source: Listing 16.2.9.1 - Vital signs Program: Tables\k343-vs-tbl.sas



Table 14.3.5.2 - Descriptive statistics of vital signs at screening and end of study - Safety set

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Diastolic Blood Pressure [mmHg] | End of Study | N | nn |
| | | Mean | xxx.x |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Heart Rate [beats/min] | Screening | N | nn |
| | 50000000 | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Heart Rate [beats/min] | End of Study | N | nn |
| , | • | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |

Note: End of Study = Visit 4 - Follow-up or early termination visit

Source: Listing 16.2.9.1 - Vital signs Program: Tables\k343-vs-tbl.sas



Table 14.3.5.3 - Descriptive statistics of vital signs during the study - Safety set

| | | | Safety S | Set |
|---|---|---|---|---|
| Parameter | Time Point | Statistics | Chloroprocaine 3% ocular gel N=XX | Placebo<br>N=XX |
| Systolic Blood Pressure [mmHg] | Pre-dose | N | nn | nn |
| Systone Blood Fressure [mmrg] | 110 0000 | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | XXX.X |
| | | Max | XXX | XXX |
| | | 111411 | | |
| Systolic Blood Pressure [mmHg] | Post-dose | N | nn | nn |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | XXX.X |
| | | Max | XXX | XXX |
| Diastolic Blood Pressure [mmHg] | Pre-dose | N | nn | nn |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | XXX.X |
| | | Max | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.1 - Vital signs Program: Tables\k343-vs-tbl.sas



Table 14.3.5.3 - Descriptive statistics of vital signs during the study - Safety set

| | | | Safety S | Set |
|---|---|---|---|---|
| Parameter | Time Point | Statistics | Chloroprocaine 3%<br>ocular gel<br>N=XX | Placebo<br>N=XX |
| Diastolic Blood Pressure [mmHg] | Post-dose | N | nn | nn |
| | 1 000 0000 | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | XXX.X |
| | | Max | XXX | XXX |
| Heart Rate [beats/min] | Pre-dose | N | nn | nn |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | XXX.X |
| | | Max | XXX | XXX |
| Heart Rate [beats/min] | Post-dose | N | nn | nn |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | XXX.X |
| | | Max | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.1 - Vital signs Program: Tables\k343-vs-tbl.sas



# Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

### Safety Set (N=XX)

| | | | | Right Eye | | Left Eye |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Burning [mm] | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | xx.x | | xx.x | |
| | | Max | xxx | | XXX | |
| Burning [mm] | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | xx.x | | xx.x | |
| | | CV% | xx.x | | xx.x | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | xx.x | |
| | | Max | xxx | | xxx | |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

### Safety Set (N=XX)

| | | | | Right Eye | | Left Eye |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Burning [mm] | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |
| Burning [mm] | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| Burning [mm] | visit 4 - 1 ollow-up | | | | | |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

### Safety Set (N=XX)

| | | | | Right Eye | | Left Eye |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Stinging [mm] | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | xx.x | | xx.x | |
| | | Max | XXX | | xxx | |
| Stinging [mm] | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | xx.x | | xx.x | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | xx.x | | xx.x | |
| | | Max | xxx | | xxx | |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

### Safety Set (N=XX)

| | | | | Right Eye | | Left Eye |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Stinging [mm] | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |
| Stinging [mm] | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | • | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | xx.x | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | xx.x | XX.X |
| | | Max | xxx | XXX | xxx | XXX |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

 $Program: Tables \backslash k343\text{-}qs\text{-}tbl.sas$ 



Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

### Safety Set (N=XX)

| | | | | Right Eye | | Left Eye |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Itching [mm] | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | xx.x | |
| | | Max | xxx | | XXX | |
| Itching [mm] | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | xx.x | | xx.x | |
| | | Max | XXX | | xxx | |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

### Safety Set (N=XX)

| | | | Right Eye | | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Itching [mm] | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |
| Itching [mm] | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | xx.x | XX.X | xx.x | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

### Safety Set (N=XX)

| | | | Right Eye | | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Foreign Body Sensation [mm] | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | XXX | | XXX | |
| Foreign Body Sensation [mm] | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | xx.x | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | XXX | | XXX | |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

### Safety Set (N=XX)

| | | | Right Eye | | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Foreign Body Sensation [mm] | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | xxx | XXX |
| Foreign Body Sensation [mm] | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | xxx | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | xxx | XXX |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



### Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

**Investigational Product: Placebo** 

### Safety Set (N=XX)

| | | | Right Eye | | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Burning [mm] | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | xxx | | XXX | |
| Burning [mm] | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | xx.x | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | xxx | | xxx | |

Note: Subjects are summarised according to the product they actually received \_

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

**Investigational Product: Placebo** 

#### Safety Set (N=XX)

| | | | | Suicty Set | Surety Set (11 7221) | |
|---|---|---|---|---|---|---|
| | | | | Right Eye | Left Eye | |
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | <b>Change from Baseline</b> |
| Burning [mm] | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | xxx | XXX | xxx |
| Burning [mm] | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | xxx | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received \_

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



### Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

**Investigational Product: Placebo** 

### Safety Set (N=XX)

| | | | Right Eye | | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Stinging [mm] | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | XXX | | XXX | |
| Stinging [mm] | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | XXX | | xxx | |

Note: Subjects are summarised according to the product they actually received \_

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



### Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

**Investigational Product: Placebo** 

### Safety Set (N=XX)

| | | | Right Eye | | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Stinging [mm] | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | xxx | XXX | XXX | XXX |
| Stinging [mm] | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | xx.x | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | xxx | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received \_

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

**Investigational Product: Placebo** 

### Safety Set (N=XX)

| | | | Right Eye | | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Itching [mm] | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | XXX | | XXX | |
| Itching [mm] | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | xx.x | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | xxx | | XXX | |

Note: Subjects are summarised according to the product they actually received \_

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

**Investigational Product: Placebo** 

### Safety Set (N=XX)

| | | | Right Eye | | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Itching [mm] | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |
| Itching [mm] | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received \_

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



### Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

**Investigational Product: Placebo** 

### Safety Set (N=XX)

| | | | Right Eye | | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Foreign Body Sensation [mm] | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | xx.x | | XX.X | |
| | | Max | XXX | | xxx | |
| Foreign Body Sensation [mm] | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | XXX | | xxx | |

Note: Subjects are summarised according to the product they actually received \_

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



### Table 14.3.5.4 - Descriptive statistics of ocular symptoms - Safety set

**Investigational Product: Placebo** 

#### Safety Set (N=XX)

| | | | Salety Set (11-AA) | | | |
|---|---|---|---|---|---|---|
| | | | Right Eye | | Left Eye | |
| Parameter | Visit | <b>Statistics</b> | Value | Change from Baseline | Value | Change from Baseline |
| Foreign Body Sensation [mm] | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | xxx | xxx | xxx | xxx |
| Foreign Body Sensation [mm] | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | • | Mean | xx.x | XX.X | XX.X | XX.X |
| | | SD | xx.x | XX.X | XX.X | XX.X |
| | | CV% | xx.x | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | xx.x | XX.X | XX.X | XX.X |
| | | Max | xxx | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received \_

Baseline: Pre-dose assessments

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



## Table 14.3.5.5 - Wilcoxon Rank Sum Test on changes from baseline in Ocular Symptoms - Safety set

# **Change from Baseline in Burning**

| | | Rigl | nt eye | Left | Left eye |
|---|---|---|---|---|---|
| Visit | Comparison | Wilcoxon<br>Rank-Sum<br>Statistics | Wilcoxon<br>Rank-Sum<br>p-value | Wilcoxon<br>Rank-Sum<br>Statistics | Wilcoxon<br>Rank-Sum<br>p-value |
| Visit 2 - Post-dose | Chloroprocaine 3% ocular gel vs. Placebo | xx.x | x.xxxx | xx.x | x.xxxx |
| Visit 4 - Follow-up | Chloroprocaine 3% ocular gel vs. Placebo | XX.X | x.xxxx | xx.x | x.xxxx |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessment

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas


## Table 14.3.5.5 - Wilcoxon Rank Sum Test on changes from baseline in Ocular Symptoms - Safety set

# **Change from Baseline in Stinging**

| | | Rigl | nt eye | Left eye | |
|---|---|---|---|---|---|
| Visit | Comparison | Wilcoxon<br>Rank-Sum<br>Statistics | Wilcoxon<br>Rank-Sum<br>p-value | Wilcoxon<br>Rank-Sum<br>Statistics | Wilcoxon<br>Rank-Sum<br>p-value |
| Visit 2 - Post-dose | Chloroprocaine 3% ocular gel vs. Placebo | xx.x | x.xxxx | xx.x | x.xxxx |
| Visit 4 - Follow-up | Chloroprocaine 3% ocular gel vs. Placebo | XX.X | x.xxxx | xx.x | x.xxxx |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessment

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



## Table 14.3.5.5 - Wilcoxon Rank Sum Test on changes from baseline in Ocular Symptoms - Safety set

# **Change from Baseline in Itching**

| | | Rigl | nt eye | Left eye | |
|---|---|---|---|---|---|
| Visit | Comparison | Wilcoxon<br>Rank-Sum<br>Statistics | Wilcoxon<br>Rank-Sum<br>p-value | Wilcoxon<br>Rank-Sum<br>Statistics | Wilcoxon<br>Rank-Sum<br>p-value |
| Visit 2 - Post-dose | Chloroprocaine 3% ocular gel vs. Placebo | xx.x | x.xxxx | xx.x | x.xxxx |
| Visit 4 - Follow-up | Chloroprocaine 3% ocular gel vs. Placebo | XX.X | x.xxxx | xx.x | x.xxxx |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessment

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



## Table 14.3.5.5 - Wilcoxon Rank Sum Test on changes from baseline in Ocular Symptoms - Safety set

## **Change from Baseline in Foreign Body Sensation**

| | | Rigl | nt eye | Left eye | |
|---|---|---|---|---|---|
| Visit | Comparison | Wilcoxon<br>Rank-Sum<br>Statistics | Wilcoxon<br>Rank-Sum<br>p-value | Wilcoxon<br>Rank-Sum<br>Statistics | Wilcoxon<br>Rank-Sum<br>p-value |
| Visit 2 - Post-dose | Chloroprocaine 3% ocular gel vs. Placebo | xx.x | x.xxxx | XX.X | x.xxxx |
| Visit 4 - Follow-up | Chloroprocaine 3% ocular gel vs. Placebo | XX.X | x.xxxx | xx.x | x.xxxx |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessment

Source: Listing 16.2.9.2 - Ocular symptoms

Program: Tables\k343-qs-tbl.sas



## Table 14.3.5.6 - Descriptive statistics of visual Acuity - Safety set

# Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | | Safety Se | Safety Set (N-AA) |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Visual Acuity Score 1 | Screening | N | nn | nn |
| | | Mean | x.xx | x.xx |
| | | SD | x.xx | x.xx |
| | | CV% | x.xx | x.xx |
| | | Min | X.X | x.x |
| | | Median | X.XX | x.xx |
| | | Max | X.X | X.X |
| Visual Acuity Score <sup>1</sup> | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | x.xx | x.xx |
| | | SD | x.xx | x.xx |
| | | CV% | x.xx | x.xx |
| | | Min | x.x | X.X |
| | | Median | X.XX | x.xx |
| | | Max | X.X | x.x |

Note: Subjects are summarised according to the product they actually received

Note 1: Visual Acuity Score not always evaluated as best corrected, see source listing for details

Source: Listing 16.2.9.3 - Visual acuity

Program: Tables\k343-qs-tbl.sas



## Table 14.3.5.6 - Descriptive statistics of visual Acuity - Safety set

**Investigational Product: Placebo** 

#### Safety Set (N=XX)

| | | | Safety Set (N=XX) | |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Visual Acuity Score 1 | Screening | N | nn | nn |
| | | Mean | X.XX | x.xx |
| | | SD | X.XX | x.xx |
| | | CV% | x.xx | x.xx |
| | | Min | X.X | X.X |
| | | Median | x.xx | x.xx |
| | | Max | X.X | x.x |
| Visual Acuity Score 1 | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | x.xx | x.xx |
| | | SD | X.XX | x.xx |
| | | CV% | X.XX | x.xx |
| | | Min | X.X | X.X |
| | | Median | X.XX | x.xx |
| | | Max | X.X | x.x |

Note: Subjects are summarised according to the product they actually received

Note 1: Visual Acuity Score not always evaluated as best corrected, see source listing for details

Source: Listing 16.2.9.3 - Visual acuity

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

## Safety Set (N=XX)

| | | Right Eye | | | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Conjunctival redness | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | xxx | | xxx | |
| Conjunctival redness | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | xxx | | xxx | |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

 $Program: Tables \backslash k343\text{-}qs\text{-}tbl.sas$ 



# Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | | Disk For | | | |
|---|---|---|---|---|---|---|
| | | | | Right Eye | | Left Eye |
| Parameter | Visit | <b>Statistics</b> | Value | Change from Baseline | Value | Change from Baseline |
| Conjunctival redness | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | xxx | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | xxx | xxx | xxx | xxx |
| Conjunctival redness | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | xx.x | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | xx.x | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | xxx | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

 $Program: Tables \backslash k343\text{-}qs\text{-}tbl.sas$ 



# Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

## Safety Set (N=XX)

| | | | Right Eye | | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Anterior chamber flare | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | xxx | | xxx | |
| Anterior chamber flare | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | xx.x | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | xx.x | |
| | | Max | xxx | | xxx | |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | Suitely Set (1. 1212) | | | | |
|---|---|---|---|---|---|---|
| | | | | Right Eye | Left Eye | |
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | <b>Change from Baseline</b> |
| Anterior chamber flare | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | xxx | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | xxx | xxx | XXX | xxx |
| Anterior chamber flare | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | xx.x | XX.X | XX.X | XX.X |
| | | SD | xx.x | XX.X | XX.X | XX.X |
| | | CV% | xx.x | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | xxx | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

 $Program: Tables \backslash k343\text{-}qs\text{-}tbl.sas$ 



# Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

## Safety Set (N=XX)

| | | | Right Eye | | | Left Eye |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Conjunctival chemosis | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | XXX | | XXX | |
| Conjunctival chemosis | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | XXX | | XXX | |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

## Safety Set (N=XX)

| | | | | Right Eye | | Left Eye |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Conjunctival chemosis | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | xxx | XXX |
| | 77 5 A 77 H | 3.7 | | | | |
| Conjunctival chemosis | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | xxx | XXX | xxx | XXX |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

 $Program: Tables \backslash k343\text{-}qs\text{-}tbl.sas$ 



# Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

## Safety Set (N=XX)

| | Right Eye | | | Left Eye | | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Eyelid swelling | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | XXX | | XXX | |
| Eyelid swelling | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | xx.x | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | xxx | | xxx | |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | | | Right Eye | | Left Eye |
|---|---|---|---|---|---|---|
| Parameter | Visit | <b>Statistics</b> | Value | Change from Baseline | Value | Change from Baseline |
| Eyelid swelling | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | xxx | xxx | XXX | XXX |
| Eyelid swelling | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | xx.x | XX.X | XX.X | XX.X |
| | | SD | xx.x | XX.X | XX.X | XX.X |
| | | CV% | xx.x | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | xxx | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

Program: Tables\k343-qs-tbl.sas



## Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

**Investigational Product: Placebo** 

## Safety Set (N=XX)

| | | | | Right Eye | | Left Eye |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Conjunctival redness | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | xx.x | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | xx.x | | XX.X | |
| | | Max | XXX | | xxx | |
| Conjunctival redness | Visit 2 - Pre-dose | N | nn | | nn | |
| • | | Mean | xx.x | | XX.X | |
| | | SD | xx.x | | XX.X | |
| | | CV% | xx.x | | XX.X | |
| | | Min | XXX | | xxx | |
| | | Median | xx.x | | XX.X | |
| | | Max | XXX | | xxx | |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

Program: Tables\k343-qs-tbl.sas



## Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

**Investigational Product: Placebo** 

## Safety Set (N=XX)

| | | | | Right Eye | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | <b>Change from Baseline</b> |
| Conjunctival redness | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | xxx |
| Conjunctival redness | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | xx.x | XX.X | XX.X | XX.X |
| | | SD | xx.x | XX.X | XX.X | XX.X |
| | | CV% | xx.x | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

Program: Tables\k343-qs-tbl.sas



## Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

**Investigational Product: Placebo** 

## Safety Set (N=XX)

| | | | Dight Fue | | | |
|---|---|---|---|---|---|---|
| | | | | Right Eye | | Left Eye |
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Anterior chamber flare | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | xxx | | xxx | |
| Anterior chamber flare | Visit 2 - Pre-dose | N | nn | | nn | |
| Anterior chamber hare | VISIT 2 - I Te-dose | | 1111 | | 1111 | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | XXX | | XXX | |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

 $Program: Tables \backslash k343\text{-}qs\text{-}tbl.sas$ 



Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

**Investigational Product: Placebo** 

## Safety Set (N=XX)

| | | | | Right Eye | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Anterior chamber flare | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | xxx | XXX | XXX | XXX |
| Anterior chamber flare | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

Program: Tables\k343-qs-tbl.sas



## Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

**Investigational Product: Placebo** 

## Safety Set (N=XX)

| | | Dight Evo | | | | I . & E |
|---|---|---|---|---|---|---|
| | | | | Right Eye | | Left Eye |
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Conjunctival chemosis | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | xxx | | xxx | |
| Conjunctival chemosis | Visit 2 - Pre-dose | N | nn | | nn | |
| • | | Mean | xx.x | | XX.X | |
| | | SD | xx.x | | XX.X | |
| | | CV% | xx.x | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | xx.x | | XX.X | |
| | | Max | XXX | | XXX | |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

 $Program: Tables \backslash k343\text{-}qs\text{-}tbl.sas$ 



## Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

**Investigational Product: Placebo** 

## Safety Set (N=XX)

| | | | | Right Eye | Left Eye | |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | <b>Change from Baseline</b> |
| Conjunctival chemosis | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | xx.x | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | xxx | XXX | XXX | xxx |
| Conjunctival chemosis | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | xx.x | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | xx.x | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

Program: Tables\k343-qs-tbl.sas



## Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

**Investigational Product: Placebo** 

## Safety Set (N=XX)

| | | survey set (i v illi) | | | | |
|---|---|---|---|---|---|---|
| | | | | Right Eye | | Left Eye |
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | <b>Change from Baseline</b> |
| Eyelid swelling | Screening | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | XX.X | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | xxx | | xxx | |
| Eyelid swelling | Visit 2 - Pre-dose | N | nn | | nn | |
| | | Mean | XX.X | | XX.X | |
| | | SD | XX.X | | xx.x | |
| | | CV% | XX.X | | XX.X | |
| | | Min | XXX | | XXX | |
| | | Median | XX.X | | XX.X | |
| | | Max | XXX | | XXX | |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

Program: Tables\k343-qs-tbl.sas



## Table 14.3.5.7 - Descriptive statistics of slit lamp examination - Safety set

**Investigational Product: Placebo** 

## Safety Set (N=XX)

| | | | | Right Eye | , | Left Eye |
|---|---|---|---|---|---|---|
| Parameter | Visit | Statistics | Value | Change from Baseline | Value | Change from Baseline |
| Eyelid swelling | Visit 2 - Post-dose | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |
| Eyelid swelling | Visit 4 - Follow-up | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XXX | XXX | XXX | XXX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XXX | XXX | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Baseline: Pre-dose assessments

Source: Listing 16.2.9.4 - Slit lamp examination

 $Program: Tables \backslash k343\text{-}qs\text{-}tbl.sas$ 



Table 14.3.5.8 - Descriptive statistics of corneal fluorescein staining - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | | Safety Set (N=XX) | |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Central Cornea | Screening | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | X |
| Central Cornea | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.5 - Corneal fluorescein staining

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.8 - Descriptive statistics of corneal fluorescein staining - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | Safety Set (N=XX) | | |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Superior Cornea | Screening | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | X |
| Superior Cornea | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.5 - Corneal fluorescein staining

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.8 - Descriptive statistics of corneal fluorescein staining - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | Safety Set (N=XX) | | |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Inferior Cornea | Screening | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | X |
| Inferior Cornea | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.5 - Corneal fluorescein staining

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.8 - Descriptive statistics of corneal fluorescein staining - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | | Salety St | et (IN-AA) |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Nasal Cornea | Screening | N | nn | nn |
| | | Mean | X.X | X.X |
| | | SD | X.X | X.X |
| | | CV% | X.X | X.X |
| | | Min | X | x |
| | | Median | X.X | X.X |
| | | Max | x | X |
| Nasal Cornea | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | X.X |
| | | SD | X.X | X.X |
| | | CV% | X.X | X.X |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | X |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.5 - Corneal fluorescein staining

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.8 - Descriptive statistics of corneal fluorescein staining - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | | Safety Se | (N=XX) |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Temporal Cornea | Screening | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | X.X |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | X |
| Temporal Cornea | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.5 - Corneal fluorescein staining

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.8 - Descriptive statistics of corneal fluorescein staining - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | | Safety Set (N=XX) | |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Total Score | Screening | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | X |
| Total Score | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.5 - Corneal fluorescein staining

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.8 - Descriptive statistics of corneal fluorescein staining - Safety set

**Investigational Product: Placebo** 

Safety Set (N=XX)

| | | | Safety Set (N=XX) | |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Central Cornea | Screening | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |
| Central Cornea | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.5 - Corneal fluorescein staining

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.8 - Descriptive statistics of corneal fluorescein staining - Safety set

# **Investigational Product: Placebo**

#### Safety Set (N=XX)

| | | | Safety Set (N=XX) | |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| | | | | - |
| Superior Cornea | Screening | N | nn | nn |
| | | Mean | X.X | X.X |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |
| Superior Cornea | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.5 - Corneal fluorescein staining

Program: Tables\k343-qs-tbl.sas



Table 14.3.5.8 - Descriptive statistics of corneal fluorescein staining - Safety set

**Investigational Product: Placebo** 

#### Safety Set (N=XX)

| | | | Safety Se | et (N=XX) |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Inferior Cornea | Screening | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | X |
| Inferior Cornea | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.5 - Corneal fluorescein staining

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.8 - Descriptive statistics of corneal fluorescein staining - Safety set

# **Investigational Product: Placebo**

#### Safety Set (N=XX)

| | | Safety Set (N=XX) | | |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Nasal Cornea | Screening | N | nn | nn |
| | | Mean | X.X | X.X |
| | | SD | X.X | X.X |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |
| Nasal Cornea | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.5 - Corneal fluorescein staining

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.8 - Descriptive statistics of corneal fluorescein staining - Safety set

# **Investigational Product: Placebo**

#### Safety Set (N=XX)

| | | | Safety Set (N=XX) | |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Temporal Cornea | Screening | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |
| Temporal Cornea | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.5 - Corneal fluorescein staining

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.8 - Descriptive statistics of corneal fluorescein staining - Safety set

# **Investigational Product: Placebo**

#### Safety Set (N=XX)

| | | Safety Set (N=XX) | | |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Total Score | Screening | N | nn | nn |
| | | Mean | X.X | X.X |
| | | SD | X.X | X.X |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |
| Total Score | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | X.X |
| | | SD | X.X | X.X |
| | | CV% | X.X | x.x |
| | | Min | X | x |
| | | Median | X.X | x.x |
| | | Max | X | x |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.5 - Corneal fluorescein staining

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.9 - Descriptive statistics of fundus ophthalmoscopy - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | | Saicty St | λ (11- <b>/λ/λ</b> ) |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Vitreous | Screening | N | nn | nn |
| · Aleccus | Sercening | Mean | X.X | X.X |
| | | SD | X.X | X.X |
| | | CV% | X.X | X.X |
| | | Min | X | X |
| | | Median | X.X | X.X |
| | | Max | X | X |
| Vitreous | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | X.X |
| | | SD | X.X | X.X |
| | | CV% | X.X | X.X |
| | | Min | X | X |
| | | Median | X.X | X.X |
| | | Max | X | X |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.6 - Fundus ophthalmoscopy

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.9 - Descriptive statistics of fundus ophthalmoscopy - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | Salety Set (N-AA) | | |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Macula, (Peripheral) Retina and Optic Nerve Head | Screening | N | nn | nn |
| Macuia, (1 empheral) Retina and Optic Nerve fread | Screening | | nn | |
| | | Mean | X.X | X.X |
| | | SD | X.X | x.x |
| | | CV% | X.X | x.x |
| | | Min | X | X |
| | | Median | X.X | X.X |
| | | Max | X | X |
| Macula, (Peripheral) Retina and Optic Nerve Head | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | X.X |
| | | CV% | X.X | X.X |
| | | Min | X | X |
| | | Median | X.X | X.X |
| | | Max | X | X |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.6 - Fundus ophthalmoscopy

Program: Tables\k343-qs-tbl.sas



## Table 14.3.5.9 - Descriptive statistics of fundus ophthalmoscopy - Safety set

**Investigational Product: Placebo** 

#### Safety Set (N=XX)

| | | | Safety Se | Safety Set (N=XX) |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Vitreous | Screening | N | nn | nn |
| | | Mean | X.X | X.X |
| | | SD | X.X | X.X |
| | | CV% | X.X | X.X |
| | | Min | X | X |
| | | Median | X.X | X.X |
| | | Max | X | X |
| Vitreous | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | X.X |
| | | SD | X.X | X.X |
| | | CV% | X.X | X.X |
| | | Min | X | X |
| | | Median | X.X | X.X |
| | | Max | X | X |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.6 - Fundus ophthalmoscopy

Program: Tables\k343-qs-tbl.sas


#### Table 14.3.5.9 - Descriptive statistics of fundus ophthalmoscopy - Safety set

**Investigational Product: Placebo** 

#### Safety Set (N=XX)

| | | | Safety Se | t (N=XX) |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Macula, (Peripheral) Retina and Optic Nerve Head | Screening | N | nn | nn |
| | | Mean | X.X | x.x |
| | | SD | X.X | X.X |
| | | CV% | X.X | X.X |
| | | Min | X | X |
| | | Median | X.X | X.X |
| | | Max | x | X |
| Macula, (Peripheral) Retina and Optic Nerve Head | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | X.X | X.X |
| | | SD | X.X | X.X |
| | | CV% | X.X | X.X |
| | | Min | X | X |
| | | Median | X.X | X.X |
| | | Max | X | X |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.6 - Fundus ophthalmoscopy

Program: Tables\k343-qs-tbl.sas



# Table 14.3.5.10 - Descriptive statistics of intraocular pressure - Safety set

Investigational Product: Chloroprocaine 3% ocular gel

#### Safety Set (N=XX)

| | | | Safety Set (N=XX) | |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Intraocular pressure [mmHg] | Screening | N | nn | nn |
| | | Mean | xxx.x | XXX.X |
| | | SD | xxx.x | xxx.x |
| | | CV% | xxx.x | xxx.x |
| | | Min | xxx | xxx |
| | | Median | xxx.x | xxx.x |
| | | Max | XXX | xxx |
| Intraocular pressure [mmHg] | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | xxx.x | xxx.x |
| | | SD | xxx.x | xxx.x |
| | | CV% | XXX.X | xxx.x |
| | | Min | xxx | xxx |
| | | Median | XXX.X | xxx.x |
| | | Max | XXX | xxx |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.7 - Intraocular pressure

Program: Tables $\k343$ -qs-tbl.sas



# Table 14.3.5.10 - Descriptive statistics of intraocular pressure - Safety set

**Investigational Product: Placebo** 

#### Safety Set (N=XX)

| | | | Safety Se | et (N=XX) |
|---|---|---|---|---|
| Parameter | Visit | Statistics | Right Eye<br>Value | Left Eye<br>Value |
| Intraocular pressure [mmHg] | Screening | N | nn | nn |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | xxx.x |
| | | Min | XXX | xxx |
| | | Median | XXX.X | xxx.x |
| | | Max | XXX | xxx |
| Intraocular pressure [mmHg] | Visit 4 - Follow-up | N | nn | nn |
| | | Mean | XXX.X | xxx.x |
| | | SD | XXX.X | xxx.x |
| | | CV% | XXX.X | xxx.x |
| | | Min | XXX | xxx |
| | | Median | XXX.X | xxx.x |
| | | Max | XXX | xxx |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.7 - Intraocular pressure

Program: Tables $\k343$ -qs-tbl.sas


Statistical analysis plan CRO-PK-20-343

Sponsor code CHL.3-01-2020 Chloroprocaine 3% ocular gel Final version 1.0, 20NOV20



Section 16.2 - Individual Subject Data Listings Shells

| Listing | 16.2.1.1 - | Discontinued | subjects |
|---------|------------|--------------|----------|
|---------|------------|--------------|----------|

Listing 16.2.2.1 - Protocol deviations

Listing 16.2.2.2 - Assigned and actual treatment mismatches

Listing 16.2.3.1 - Subjects excluded from safety and/or efficacy analysis

Listing 16.2.4.1 - Subjects' disposition

Listing 16.2.4.2 - Analysis sets

Listing 16.2.4.3 - Demography

Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

Listing 16.2.5.1 - Investigational products administration

Listing 16.2.6.1 - Conjunctival pinching

Listing 16.2.6.2 - Anesthesia results

Listing 16.2.7.1 - Treatment-emergent adverse events

Listing 16.2.7.2 - Pre-treatment adverse events

Listing 16.2.8.1 - Alcohol Breath Test and Pregnancy Test

Listing 16.2.9.1 - Vital signs

Listing 16.2.9.2 - Ocular symptoms

Listing 16.2.9.3 - Visual acuity

Listing 16.2.9.4 - Slit Lamp Examination

Listing 16.2.9.5 - Corneal fluorescein staining

Listing 16.2.9.6 - Fundus ophthalmoscopy

Listing 16.2.9.7 - Intraocular pressure

Listing 16.2.10.1 - Medical and surgical history

Listing 16.2.10.2 - Physical examination

Listing 16.2.10.3 - Prior and concomitant medications

Listing 16.2.10.4 - Subjects study visits

Listing 16.2.10.5 - Fertility status and contraception



**Listing 16.2.1.1 - Discontinued subjects** 

| Subject<br>ID | Last IP before discontinuation | Sex | Age<br>(years) | Last<br>visit | Time elapsed from<br>last drug<br>administration<br>(days) | Date of premature discontinuation | Primary reason for subject premature study termination |
|---|---|---|---|---|---|---|---|
| S001/001 | Chloroprocaine 3% ocular gel | M | 30 | Visit 2 | 1 | ddMMMyyyy | Withdrawal by subject |
| S003/002 | Placebo | F | 27 | Visit 3 | 2 | ddMMMyyyy | Adverse event |
| S005/004 | Placebo | M | 18 | Visit 2 | 2 | ddMMMyyyy | Physician decision |
| S007/006 | Chloroprocaine 3% ocular gel | F | 27 | Visit 1 | 2 | ddMMMyyyy | Adverse event |
| S011/010 | Placebo | M | 18 | Visit 2 | 2 | ddMMMyyyy | Physician decision |
| | | ••• | | ••• | | ••• | |

Note: Subjects are listed according to the last product they actually received before discontinuation

Program: Listings\k343-ds-lst.sas



**Listing 16.2.2.1 - Protocol deviations** 

| Subject<br>ID | Deviation<br>Number | Deviation<br>Category | | Deviation Description |
|---|---|---|---|---|
| | | | Term | |
| S001/001 | 1 | Minor | Deviation from scheduled collecting time | Pinching number 1 was collected outside the window of 20 seconds after the third drop |
| S002/002 | 1 | Minor | Deviation from scheduled assessment order | Vital signs assessment were performed after ocular symptoms |
| S007/006 | 1 | Major | Inclusion criteria violation | Inclusion criteria violation |

Program: Listings\k343-dv-lst.sas




Statistical analysis plan CRO-PK-20-343 Sponsor code CHL.3-01-2020 Chloroprocaine 3% ocular gel Final version 1.0, 20NOV20

# Listing 16.2.2.2 - Assigned and actual treatment mismatches

| Subject<br>ID | Assigned Arm | Actual Arm |
|---------------|------------------------------|------------|
| S003/002 | Chloroprocaine 3% ocular gel | Placebo |
| | <b></b> | |

Program: Listings\k343-ds-lst.sas



Listing 16.2.3.1 - Subjects excluded from safety and/or efficacy analysis

| Subject<br>ID | Sex | Age<br>(years) | Enrolled<br>Set | Safety<br>Set | Full Analysis<br>Set | Per Protocol<br>Set | Reason for the exclusion |
|---|---|---|---|---|---|---|---|
| S010/008 | F | 30 | Y | N | N | N | Lack of IP intake |
| S015/013 | F | 20 | Y | Y | Y | N | Major protocol deviations |
| | ••• | | • | • | • | | |

Program: Listings\k343-ds-lst.sas



# Listing 16.2.4.1 - Subjects' disposition

| Subject<br>ID | Date of<br>Informed | Date of Screening | Date of Randomisation | Date of IP | Completed or | Date of Study<br>Completion or | Date of<br>End of | Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|
| | Consent | | | Administration | Discontinued | Discontinuation | Participation | |
| S001/001 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Discontinued | ddMMMyyyy | ddMMMyyyy | Withdrawal by subject |
| S002/002 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Completed | ddMMMyyyy | ddMMMyyyy | |
| S005/003 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Discontinued | ddMMMyyyy | ddMMMyyyy | Adverse event |
| | | | ••• | ••• | | | ••• | |

Program: Listings\k343-ds-lst.sas



# Listing 16.2.4.2 - Analysis sets

| Subject | Planned Arm | Enrolled | Safety | <b>Full Analysis</b> | Per Protocol | Reason for the exclusion |
|---|---|---|---|---|---|---|
| ID | | Set | Set | Set | Set | |
| S001/001 | Chloroprocaine 3% ocular gel | Y | N | N | N | Lack of IP intake |
| S003/002 | Placebo | Y | Y | Y | Y | |
| | <b></b> | • | • | • | • | |

Note: Subjects are listed according to the treatment they were assigned to

Program: Listings\k343-ds-lst.sas



# **Listing 16.2.4.3 - Demography**

| Subject<br>ID | Sex | Race | Birth<br>Year | Age<br>(years) | Height<br>(cm) | Body Weight (kg) | Body Mass Index<br>(kg/m²) |
|---|---|---|---|---|---|---|---|
| S001/001 | F | White | 2001 | 19 | 170 | 55.0 | 19.0 |
| S002/002 | M | White | 1990 | 30 | 187 | 91.0 | 26.0 |
| | | | | | ••• | | ··· |

Note:Program:Listings\k343-dm-lst.sas



# Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

| Subject<br>ID | Criterion | Verbatim |
|---|---|---|
| S001/001 | Exclusion criterion 2 | Visual acuity: Best corrected visual acuity < 1/10 |
| | ••• | |

Program: Listings\k343-ie-lst.sas



#### Listing 16.2.5.1 - Investigational products administration

Investigational Product: Chloroprocaine 3% ocular gel

| Subject<br>ID | Drop<br>Nr | Scheduled<br>Time | Administration Date/time |
|---|---|---|---|
| S001/001 | 1 | First drop of the IP | ddMMMyyyy hh:mm:ss |
| S001/001 | 2 | $1 \min \pm 15$ sec after the first drop of the IP | ddMMMyyyy hh:mm:ss |
| S001/001 | 3 | $1 \min \pm 15$ sec after the second drop of the IP | ddMMMyyyy hh:mm:ss |
| ••• | <b></b> | <b></b> | |

Note: Subjects are listed according to the product they actually received

Program: Listings\k343-ex-lst.sas



# Listing 16.2.5.1 - Investigational products administration

# **Investigational Product: Placebo**

| Subject<br>ID | Drop<br>Nr | Scheduled<br>Time | Administration Date/time |
|---|---|---|---|
| S007/006 | 1 | First drop of the IP | ddMMMyyyy hh:mm:ss |
| S007/006 | 2 | $1 \min \pm 15$ sec after the first drop of the IP | ddMMMyyyy hh:mm:ss |
| S007/006 | 3 | $1 \min \pm 15$ sec after the second drop of the IP | ddMMMyyyy hh:mm:ss |

Note: Subjects are listed according to the product they actually received

Program: Listings\k343-ex-lst.sas



Listing 16.2.6.1 - Conjunctival pinching

Investigational Product: Chloroprocaine 3% ocular gel

| Subject<br>ID | Pinching<br>Nr | Scheduled<br>Time | Collection<br>Date/Time | Did the subject experienced pain? |
|---|---|---|---|---|
| S001/001 | 1 | 20 seconds after the instillation of third drop | ddMMMyyyy hh:mm:ss | Y |
| S001/001 | 2 | 40 seconds after the instillation of third drop | ddMMMyyyy hh:mm:ss | Y |
| S001/001 | 3 | 60 seconds after the instillation of third drop | ddMMMyyyy hh:mm:ss | Y |
| S001/001 | 4 | 5 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 5 | 10 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 6 | 15 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 7 | 20 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 8 | 25 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 9 | 30 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 10 | 35 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 11 | 40 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 12 | 45 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 13 | 50 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 14 | 55 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 15 | 60 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |

Note: Subjects are listed according to the product they actually received

Program: Listings\k343-eff-lst.sas



# Listing 16.2.6.1 - Conjunctival pinching

**Investigational Product: Placebo** 

| Subject<br>ID | Pinching<br>Nr | Scheduled<br>Time | Collection<br>Date/Time | Did the subject experienced pain? |
|---|---|---|---|---|
| S001/001 | 1 | 20 seconds after the instillation of third drop | ddMMMyyyy hh:mm:ss | Y |
| S001/001 | 2 | 40 seconds after the instillation of third drop | ddMMMyyyy hh:mm:ss | Y |
| S001/001 | 3 | 60 seconds after the instillation of third drop | ddMMMyyyy hh:mm:ss | Y |
| S001/001 | 4 | 5 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 5 | 10 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 6 | 15 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 7 | 20 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 8 | 25 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 9 | 30 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 10 | 35 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 11 | 40 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 12 | 45 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 13 | 50 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 14 | 55 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| S001/001 | 15 | 60 minutes after the instillation of third drop | ddMMMyyyy hh:mm:ss | N |
| | ••• | | | |

Note: Subjects are listed according to the product they actually received

Program: Listings\k343-eff-lst.sas



#### Listing 16.2.6.2 - Anesthesia results

#### **Investigational Product: Chloroprocaine 3% ocular gel**

| Subject<br>ID | Anesthesia Success <sup>1</sup> | Time to Anesthesia <sup>2</sup> (min) | Anesthesia Duration <sup>3</sup> (min) |
|---|---|---|---|
| S001/001 | Y | 5 | 25 |
| S002/002 | N | | <del></del> |
| ••• | | | <b></b> |

Note: Subjects are listed according to the product they actually received

Note 1: Anesthesia Succes is defined as full anesthesia of the ocular surface 5 minutes after administration of the investigational product

Note 2: Time to Anesthesia is defined as time of the second test, in case of two successive tests with no pain, or 5 minutes after administration of the investigational product

Note 3: Anesthesia Duration is defines as the interval between Time to Anesthesia and the time of the first test, in case of two successive tests with pain

Program:Listings\k343-eff-lst.sas




#### Listing 16.2.6.2 - Anesthesia results

#### **Investigational Product: Placebo**

| Subject<br>ID | Anesthesia Success <sup>1</sup> | Time to Anesthesia <sup>2</sup> (min) | Anesthesia Duration <sup>3</sup> (min) |
|---|---|---|---|
| S007/003 | Y | 5 | 25 |
| S012/005 | N | | |
| ••• | <b></b> | | |

Note: Subjects are listed according to the product they actually received

Note 1: Anesthesia Succes is defined as full anesthesia of the ocular surface 5 minutes after administration of the investigational product

Note 2: Time to Anesthesia is defined as time of the second test, in case of two successive tests with no pain, or 5 minutes after administration of the investigational product

Note 3: Anesthesia Duration is defines as the interval between Time to Anesthesia and the time of the first test, in case of two successive tests with pain

Program:Listings\k343-eff-lst.sas




# Listing 16.2.7.1 - Treatment-emergent adverse events

#### **Investigational Product: Chloroprocaine 3% ocular gel**

| Subject<br>ID | Adverse<br>Event<br>ID | Follow<br>Up<br>ID | , | |
|---|---|---|---|---|
| S001/001 | 1 | | Description: | Headache |
| | | | Body Area Affected: | Head |
| | | | Preferred Term <sup>1</sup> : | Headache |
| | | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | | Acknowledgment Date/Time (Day) | ddMMMyyyy hh:mm (j) |
| | | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | | Duration: | xx h xx min |
| | | | Has the Adverse Event Started After the Administration of the Study Drug? | Y |
| | | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | | Time Elapsed form Last Study Drug intake before AE: | xx h xx min |
| | | | Reasonable Possibility of a Causal Relationship with the Study Drug? | Y |
| | | | Other Causal Relationship: | |
| | | | Severity: | Mild |
| | | | Pattern: | Continuous |
| | | | Serious Adverse Event? / Seriousness criteria: | N / |
| | | | Action taken with Study Drug: | Dose not changed |
| | | | Concomitant Therapy? | Y |
| | | | Caused Study Discontinuation? | N |
| | | | Other Action Taken: | |
| | | | Outcome: | Recovered/Resolved |
| | | | Comments: | |
| | ••• | ••• | | ··· |

Note: Subjects are listed according to the product they actually received

Note 1: MedDRA version xx.x Program: Listings\k343-ae-lst.sas



# Listing 16.2.7.1 - Treatment-emergent adverse events

#### **Investigational Product: Placebo**

| Subject<br>ID | Adverse<br>Event<br>ID | Follow<br>Up<br>ID | , | |
|---|---|---|---|---|
| S001/001 | 2 | | Description: | Headache |
| | | | Body Area Affected: | Head |
| | | | Preferred Term <sup>1</sup> : | Headache |
| | | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | | Acknowledgment Date/Time (Day) | ddMMMyyyy hh:mm (j) |
| | | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | | Duration: | xx h xx min |
| | | | Has the Adverse Event Started After the Administration of the Study Drug? | Y |
| | | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | | Time Elapsed form Last Study Drug intake before AE: | xx h xx min |
| | | | Reasonable Possibility of a Causal Relationship with the Study Drug? | Y |
| | | | Other Causal Relationship: | |
| | | | Severity: | Mild |
| | | | Pattern: | Continuous |
| | | | Serious Adverse Event? / Seriousness criteria: | N / |
| | | | Action taken with Study Drug: | Dose not changed |
| | | | Concomitant Therapy? | Y |
| | | | Caused Study Discontinuation? | N |
| | | | Other Action Taken: | |
| | | | Outcome: | Recovered/Resolved |
| | | | Comments: | |

Note: Subjects are listed according to the product they actually received

Note 1: MedDRA version xx.x Program: Listings\k343-ae-lst.sas



# Listing 16.2.7.2 - Pre-treatment adverse events

| Subject<br>ID | Adverse<br>Event<br>ID | Follow<br>Up<br>ID | | |
|---|---|---|---|---|
| S001/001 | 1 | | Description: | Headache |
| | | | Body Area Affected: | Head |
| | | | Preferred Term <sup>1</sup> : | Headache |
| | | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | | Acknowledgment Date/Time (Day) | ddMMMyyyy hh:mm (j) |
| | | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | | Duration: | xx h xx min |
| | | | Has the Adverse Event Started After the Administration of the Study Drug? | Y |
| | | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | | Time Elapsed form Last Study Drug intake before AE: | xx h xx min |
| | | | Reasonable Possibility of a Causal Relationship with the Study Drug? | Y |
| | | | Other Causal Relationship: | |
| | | | Severity: | Mild |
| | | | Pattern: | Continuous |
| | | | Serious Adverse Event? / Seriousness criteria: | N / |
| | | | Action taken with Study Drug: | Dose not changed |
| | | | Concomitant Therapy? | Y |
| | | | Caused Study Discontinuation? | N |
| | | | Other Action Taken: | |
| | | | Outcome: | Recovered/Resolved |
| | | | Comments: | |
| ••• | | | | |

Note 1: MedDRA version xx.x Program: Listings\k343-ae-lst.sas



# **Listing 16.2.8.1 - Alcohol Breath Test and Pregnancy Test**

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value | Reference Value | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Pregnancy Test | Negative | Negative | N |
| S001/001 | Visit 2 - Day 1 | ddMMMyyyy hh:mm | Alcohol Breath Test | Negative | Negative | N |
| ••• | | | | | | ••• |

Program: Listings\k343-lb-lst.sas



# Listing 16.2.9.1 - Vital signs

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| | | | | ••• | | |

Note 1: N=Normal, H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k343-vs-lst.sas



Listing 16.2.9.2 - Ocular symptoms

Investigational Product: Chloroprocaine 3% ocular gel

| | | | | Righ | nt Eye | Lef | t Eye |
|---|---|---|---|---|---|---|---|
| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Parameter | Value | Change<br>from<br>Baseline | Value | Change<br>from<br>Baseline |
| S001/001 | Screening | ddMMMyyyy hh:mm | Burning [mm] | XX | | XX | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Stinging [mm] | XX | | XX | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Itching [mm] | XX | | XX | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Foreign Body Sensation [mm] | XX | | XX | |
| S001/001 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Burning [mm] | XX | | XX | |
| S001/001 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Stinging [mm] | XX | | XX | |
| S001/001 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Itching [mm] | XX | | XX | |
| S001/001 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Foreign Body Sensation [mm] | XX | | XX | |
| S001/001 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Burning [mm] | XX | XX | XX | XX |
| S001/001 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Stinging [mm] | XX | XX | XX | XX |
| S001/001 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Itching [mm] | XX | XX | XX | XX |
| S001/001 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Foreign Body Sensation [mm] | XX | XX | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Burning [mm] | XX | XX | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Stinging [mm] | XX | XX | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Itching [mm] | XX | XX | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Foreign Body Sensation [mm] | XX | XX | XX | XX |

Note: Subjects are listed according to the product they actually received

Baseline: Pre-dose assessments Program: Listings\k343-qs-lst.sas



# Listing 16.2.9.2 - Ocular symptoms

**Investigational Product: Placebo** 

| | Time Assessment Parameter Point Date/Time | | | Right Eye | | Left Eye | |
|---|---|---|---|---|---|---|---|
| Subject<br>ID | | | Value | Change<br>from<br>Baseline | Value | Change<br>from<br>Baseline | |
| S007/006 | Screening | ddMMMyyyy hh:mm | Burning [mm] | XX | | XX | |
| S007/006 | Screening | ddMMMyyyy hh:mm | Stinging [mm] | XX | | XX | |
| S007/006 | Screening | ddMMMyyyy hh:mm | Itching [mm] | XX | | XX | |
| S007/006 | Screening | ddMMMyyyy hh:mm | Foreign Body Sensation [mm] | XX | | XX | |
| S007/006 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Burning [mm] | XX | | XX | |
| S007/006 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Stinging [mm] | XX | XX | | |
| S007/006 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Itching [mm] | XX | xx xx | | |
| S007/006 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Foreign Body Sensation [mm] | XX | | XX | |
| S007/006 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Burning [mm] | XX | XX | XX | XX |
| S007/006 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Stinging [mm] | XX | XX | XX | XX |
| S007/006 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Itching [mm] | XX | XX | XX | XX |
| S007/006 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Foreign Body Sensation [mm] | XX | XX | XX | XX |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Burning [mm] | XX | XX | XX | XX |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Stinging [mm] | XX | XX | XX | XX |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Itching [mm] | XX | XX | XX | XX |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Foreign Body Sensation [mm] | XX | XX | XX | XX |

Note: Subjects are listed according to the product they actually received

Baseline: Pre-dose assessments Program: Listings\k343-qs-lst.sas



# Listing 16.2.9.3 - Visual acuity

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Right eye<br>Value | Left eye<br>Value | Comment |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Visual Acuity Score | X.X | X.X | |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Visual Acuity Score | X.X | X.X | |
| S007/006 | Screening | ddMMMyyyy hh:mm | Visual Acuity Score | X.X | X.X | |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Visual Acuity Score | X.X | X.X | |
| ••• | ••• | ••• | ••• | ••• | ••• | |

Program: Listings\k343-qs-lst.sas



# **Listing 16.2.9.4 - Slit Lamp Examination**

Investigational Product: Chloroprocaine 3% ocular gel

| | Time Assessment Parameter Point Date/Time | | | Rigl | ht Eye | Eye Lef | |
|---|---|---|---|---|---|---|---|
| Subject<br>ID | | | Parameter | Value | Change<br>from<br>Baseline | Value | Change<br>from<br>Baseline |
| S001/001 | Screening | ddMMMyyyy hh:mm | Conjunctival redness | XX | | XX | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Anterior chamber flare | XX | | XX | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Conjunctival chemosis | XX | | XX | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Eyelid swelling | XX | | XX | |
| S001/001 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Conjunctival redness | XX | | XX | |
| S001/001 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Anterior chamber flare | XX | XX | | |
| S001/001 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Conjunctival chemosis | XX | XX | | |
| S001/001 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Eyelid swelling | XX | | XX | |
| S001/001 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Conjunctival redness | XX | XX | XX | XX |
| S001/001 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Anterior chamber flare | XX | XX | XX | XX |
| S001/001 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Conjunctival chemosis | XX | XX | XX | XX |
| S001/001 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Eyelid swelling | XX | XX | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Conjunctival redness | XX | XX | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Anterior chamber flare | XX | XX | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Conjunctival chemosis | XX | XX | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Eyelid swelling | xx | XX | XX | XX |

Note: Subjects are listed according to the product they actually received

Baseline: Pre-dose assessments Program: Listings\k343-qs-lst.sas



# **Listing 16.2.9.4 - Slit Lamp Examination**

**Investigational Product: Placebo** 

| | | | | Rigl | nt Eye | Left Eye | |
|---|---|---|---|---|---|---|---|
| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Parameter | Value | Change<br>from<br>Baseline | Value | Change<br>from<br>Baseline |
| S007/006 | Screening | ddMMMyyyy hh:mm | Conjunctival redness | XX | | XX | |
| S007/006 | Screening | ddMMMyyyy hh:mm | Anterior chamber flare | XX | | XX | |
| S007/006 | Screening | ddMMMyyyy hh:mm | Conjunctival chemosis | XX | | XX | |
| S007/006 | Screening | ddMMMyyyy hh:mm | Eyelid swelling | XX | | XX | |
| S007/006 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Conjunctival redness | XX | | XX | |
| S007/006 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Anterior chamber flare | XX | XX | | |
| S007/006 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Conjunctival chemosis | XX | | XX | |
| S007/006 | Visit 2 - Pre-dose | ddMMMyyyy hh:mm | Eyelid swelling | XX | | XX | |
| S007/006 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Conjunctival redness | XX | XX | XX | XX |
| S007/006 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Anterior chamber flare | XX | XX | XX | XX |
| S007/006 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Conjunctival chemosis | XX | XX | XX | XX |
| S007/006 | Visit 2 - Post-dose | ddMMMyyyy hh:mm | Eyelid swelling | XX | XX | XX | XX |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Conjunctival redness | XX | XX | XX | XX |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Anterior chamber flare | XX | XX | XX | XX |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Conjunctival chemosis | XX | XX | XX | XX |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Eyelid swelling | XX | XX | XX | XX |

Note: Subjects are listed according to the product they actually received

Baseline: Pre-dose assessments Program: Listings\k343-qs-lst.sas



**Listing 16.2.9.5 - Corneal fluorescein staining** 

| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Parameter | Right eye<br>Value | Left eye<br>Value |
|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Central Cornea | xx | XX |
| S001/001 | Screening | ddMMMyyyy hh:mm | Superior Cornea | XX | XX |
| S001/001 | Screening | ddMMMyyyy hh:mm | Inferior Cornea | XX | XX |
| S001/001 | Screening | ddMMMyyyy hh:mm | Nasal Cornea | XX | XX |
| S001/001 | Screening | ddMMMyyyy hh:mm | Temporal Cornea | XX | XX |
| S001/001 | Screening | ddMMMyyyy hh:mm | Total Score | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Central Cornea | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Superior Cornea | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Inferior Cornea | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Nasal Cornea | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Temporal Cornea | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Total Score | XX | XX |
| S007/006 | Screening | ddMMMyyyy hh:mm | Central Cornea | XX | XX |
| S007/006 | Screening | ddMMMyyyy hh:mm | Superior Cornea | XX | XX |
| S007/006 | Screening | ddMMMyyyy hh:mm | Inferior Cornea | XX | XX |
| S007/006 | Screening | ddMMMyyyy hh:mm | Nasal Cornea | XX | XX |
| S007/006 | Screening | ddMMMyyyy hh:mm | Temporal Cornea | XX | XX |
| S007/006 | Screening | ddMMMyyyy hh:mm | Total Score | XX | xx |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Central Cornea | XX | xx |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Superior Cornea | XX | xx |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Inferior Cornea | XX | xx |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Nasal Cornea | XX | xx |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Temporal Cornea | XX | xx |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Total Score | XX | XX |
| ••• | | | | | |

Program: Listings\k343-qs-lst.sas



# Listing 16.2.9.6 - Fundus ophthalmoscopy

| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Parameter | Right eye<br>Value | Left eye<br>Value | Relevant<br>findings |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Vitreous | XX | XX | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Macula, (Peripheral) Retina and Optic Nerve Head | XX | XX | |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Vitreous | XX | XX | |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Macula, (Peripheral) Retina and Optic Nerve Head | XX | XX | |
| S007/006 | Screening | ddMMMyyyy hh:mm | Vitreous | XX | XX | |
| S007/006 | Screening | ddMMMyyyy hh:mm | Macula, (Peripheral) Retina and Optic Nerve Head | XX | XX | |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Vitreous | XX | XX | |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Macula, (Peripheral) Retina and Optic Nerve Head | XX | XX | |
| | | ••• | | ••• | | |

Program: Listings\k343-qs-lst.sas



# **Listing 16.2.9.7 - Intraocular pressure**

| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Parameter | Right eye<br>Value | Left eye<br>Value |
|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Intraocular Pressure [mmHg] | XX | XX |
| S001/001 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Intraocular Pressure [mmHg] | XX | XX |
| S007/006 | Screening | ddMMMyyyy hh:mm | Intraocular Pressure [mmHg] | XX | XX |
| S007/006 | Visit 4 - Follow-up | ddMMMyyyy hh:mm | Intraocular Pressure [mmHg] | XX | XX |

Program: Listings\k343-qs-lst.sas



# Listing 16.2.10.1 - Medical and surgical history

| Subject<br>ID | Category | Disease/Surgery<br>ID | | |
|---|---|---|---|---|
| S001/001 | Ocular History | M1 | Verbatim: | Strabismus |
| | | | Preferred Term 1: | Strabismus |
| | | | System Organ Class 1: | Eye disorders |
| | | | Disease Start - End Date: | 2005 - Ongoing |
| | Medical History | M1 | Verbatim: | Left shoulder luxation |
| | | | Preferred Term 1: | Joint dislocation |
| | | | System Organ Class 1: | Injury, poisoning and procedural complications |
| | | | Disease Start - End Date: | 2012 - 2012 |
| | Ocular Surgery | S1 | Verbatim: | Myopia correction |
| | | | Preferred Term 1: | Myopia correction |
| | | | System Organ Class 1: | Surgical and medical procedures |
| | | | Surgery Date: | 04NOV2007 |
| | Surgery | S1 | Verbatim: | Right knee meniscectomy |
| | | | Preferred Term 1: | Meniscus removal |
| | | | System Organ Class 1: | Surgical and medical procedures |
| | | | Surgery Date: | 04NOV1980 |
| | | ••• | | |

Note 1: MedDRA version xx.x Program: Listings\k343-mh-lst.sas



# Listing 16.2.10.2 - Physical examination

| Subject<br>ID | Time Point | Physical<br>Examination | | |
|---|---|---|---|---|
| | | Date | | |
| S001/001 | Screening | ddMMMyyyy | Investigator's Interpretation | Normal |
| | End of Study | ddMMMyyyy | Investigator's Interpretation: | Abnormal, Clinically Significant |
| | | | Clinically Significant Abnormalities: | Intraocular inflammation |
| | | | Preferred Term 1: | Eye inflammation |
| | | | System Organ Class 1: | Eye disorders |
| ••• | | | | <b></b> |

Note 1: MedDRA version xx.x Program: Listings\k343-pe-lst.sas



# Listing 16.2.10.3 - Prior and concomitant medications

| Subject<br>ID | Category | Medication ID | | |
|---|---|---|---|---|
| S001/001 | Prior | 1 | Verbatim: | Alerid |
| | | | Standardised Medication Name 1: | Alerid |
| | | | Active Ingredients 1: | Cetirizine hydrochloride |
| | | | Medication Class 1, 2: | Piperazine derivatives (R06AE) |
| | | | Indication: | Pollinosis |
| | | | Dose: | 10 mg |
| | | | Start - End Date/Time: | 2013 - Ongoing |
| | | | Frequency - Dosage Form - Route: | 1 time per day - Tablet - Oral |
| | | | Related to: | Disease M1 |
| | Concomitant | 2 | Verbatim: | Paracen |
| | | | Standardised Medication Name 1: | Paracen |
| | | | Active Ingredients 1: | Paracetamol |
| | | | Medication Class <sup>1, 2</sup> : | Anilides (N02BE) |
| | | | Indication: | Headache |
| | | | Dose: | 500 mg |
| | | | Start - End Date/Time: | 15JUN2016 19:08 - 15JUN2016 19:08 |
| | | | Frequency - Dosage Form - Route: | Once - Tablet - Oral |
| | | | Related to: | Adverse Event 1 |

Note 1: WHO Drug Dictionary Enhanced Month 1, 2020

Note 2: Anatomical Therapeutic Chemical classification, 4th level term

Program: Listings\k343-cm-lst.sas



# Listing 16.2.10.4 - Subjects study visits

| Subject<br>ID | Visit 1<br>Screening - Day -21/-1<br>Date (Day) | Visit 2<br>Day 1<br>Date (Day) | Visit 3<br>Telephone Call - Day 2<br>Date (Day) | Visit 4<br>Follow-up - Day 7±1<br>Date (Day) | Early Termination<br>Visit<br>Date (Day) |
|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy (-x) | ddMMMyyyy (x) | ddMMMyyyy (x) | ddMMMyyyy (x) | |
| S002/002 | ddMMMyyyy (-x) | ddMMMyyyy(x) | ddMMMyyyy (x) | ddMMMyyyy (x) | |
| | | | | ··· | |

Note: Program: Listings\k343-sv-lst.sas



# Listing 16.2.10.5 - Fertility status and contraception

| Subject<br>ID | Chilbearing Potential? | Non-childbearing<br>Potential<br>Status Onset | Menopausal<br>Status? | Date of<br>Menopause | Surgical<br>Sterilisation? | Surgical<br>Sterilisation<br>Date | Reliable<br>Contraceptive<br>Method Used? |
|---|---|---|---|---|---|---|---|
| S001/001 | No | ddMMMyyyy | Yes | MMMyyyy | Yes | ddMMMyyyy | |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Only female subjects are listed Program: Listings\k343-rp-lst.sas